CLINICAL TRIAL: NCT05182125
Title: A Phase 1 Clinical Trial to Evaluate the Safety and Immunogenicity of HIV-1 Vaccines Based on Chimpanzee Serotypes of Adenovirus Expressing Clade C gp140 and a CH505TF gp120 Protein Boost in Healthy, HIV- Uninfected Adult Participants
Brief Title: Phase 1 Clinical Trial to Evaluate the Safety and Immunogenicity of HIV-1 Chimp Adenovirus Vaccines Expressing Clade C gp140 & CH505TF gp120 Protein Boost in HIV-uninfected Adult.
Acronym: HVTN139
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HIV Vaccine Trials Network (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); National Institutes of Health (NIH) (NIH); Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HVTN 139; UM1AI068614 (NIH)
Record Dates: First submitted 2021-12-20; First posted 2022-01-10 (Actual); Results first posted 2024-11-27 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: HIV Infections
Keywords: HIV
MeSH Terms: conditions — HIV Infections | interventions — Product Labeling

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Part A, Group 1: AdC6-HIVgp140 (Experimental): Participants will receive 1 x 10^10 vp AdC6-HIVgp140 to be administered as two separate 1 mL IM injections into the deltoid of the non-dominant arm unless medically contraindicated at month 0.
  Interventions: Biological: AdC6-HIVgp140
- Part A, Group 2: AdC7-HIVgp140 (Experimental): Participants will receive 1 x 10^10 vp AdC7-HIVgp140 to be administered as two separate 1 mL IM injections into the deltoid of the non-dominant arm unless medically contraindicated at month 0.
  Interventions: Biological: AdC7-HIVgp140
- Part A, Group 3: Placebo (Placebo Comparator): Participants will receive placebo for AdC6-HIVgp140 or AdC7-HIVgp140 (labeled as Sodium Chloride for Injection, 0.9%) to be administered as two separate 1 mL IM injections into the deltoid of the non-dominant arm unless medically contraindicated at month 0.
  Interventions: Biological: Placebo
- Part B, Group 4: AdC6-HIVgp140 + AdC7-HIVgp140 + 400 mcg CH505TF gp120/GLA-SE (Experimental): Participants will receive 5 x 10^10 vp AdC6-HIVgp140 to be administered as two separate 1 mL IM injections into the deltoid of the non-dominant arm unless medically contraindicated at month 0.
  Then
  5 x 10^10 vp AdC7-HIVgp140 to be administered as two separate 1 mL IM injections into the deltoid of the non-dominant arm unless medically contraindicated at month 3.
  Then
  400 mcg CH505TF gp120 admixed with 10 mcg GLA-SE administered as a 1mL IM injection into either thigh unless medically contraindicated at month 6.
  Interventions: Biological: AdC6-HIVgp140; Biological: AdC7-HIVgp140; Biological: CH505TF gp120; Biological: GLA-SE (glucopyranosyl lipid A - stable emulsion; [labeled as AP 10-201])
- Part B, Group 5: AdC7-HIVgp140 + AdC6-HIVgp140 + 400 mcg CH505TF gp120/GLA-SE (Experimental): Participants will receive 5 x 10^10 vp AdC7-HIVgp140 to be administered as two separate 1 mL IM injections into the deltoid of the non-dominant arm unless medically contraindicated at month 0.
  Then
  5 x 10^10 vp AdC6-HIVgp140 to be administered as two separate 1 mL IM injections into the deltoid of the non-dominant arm unless medically contraindicated at month 3.
  Then
  400 mcg CH505TF gp120 admixed with 10 mcg GLA-SE administered as a 1mL IM injection into either thigh unless medically contraindicated at month 6.
  Interventions: Biological: AdC6-HIVgp140; Biological: AdC7-HIVgp140; Biological: CH505TF gp120; Biological: GLA-SE (glucopyranosyl lipid A - stable emulsion; [labeled as AP 10-201])
- Part B, Group 6: Placebo + Placebo + Placebo (Placebo Comparator): Participants will receive placebo for AdC6-HIVgp140and AdC7-HIVgp140 (labeled as Sodium Chloride for Injection, 0.9%) to be administered as two separate 1 mL IM injections into the deltoid of the non-dominant arm unless medically contraindicated at month 0 and 3. Placebo for CH505TF/GLA-SE (labeled as Sodium Chloride for Injection, 0.9% ) to be administered as 1 mL IM injection into either thigh at month 6.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: AdC6-HIVgp140 — The product is diluted in 2.5% Glycerol/25 mM NaCl/20 mM TRIS [tris(hydroxymethyl)aminomethane], pH 8.0 formulation buffer to a concentration of 1.2 x 10^11 vp/mL and filled at 0.3 mL for AdC6-HIVgp140 into a 2 mL Type 1 glass vial and stoppered with a gray chlorobutyl rubber stopper. The product is clear to slightly cloudy liquid, essentially free of visible particles.
  AdC6-HIVgp140 should be stored at ≤ -65°C prior to use/preparation.
  The study product is described in further detail in the Investigator's Brochure (IB).
  Arms: Part A, Group 1: AdC6-HIVgp140; Part B, Group 4: AdC6-HIVgp140 + AdC7-HIVgp140 + 400 mcg CH505TF gp120/GLA-SE; Part B, Group 5: AdC7-HIVgp140 + AdC6-HIVgp140 + 400 mcg CH505TF gp120/GLA-SE
Biological: AdC7-HIVgp140 — The products is diluted in 2.5% Glycerol/25 mM NaCl/20 mM TRIS [tris(hydroxymethyl)aminomethane], pH 8.0 formulation buffer to a concentration of 1.2 x 10^11 vp/mL and filled at 0.6 mL for AdC7-HIVgp140 into a 2 mL Type 1 glass vial and stoppered with a gray chlorobutyl rubber stopper. The product is clear to slightly cloudy liquid, essentially free of visible particles.
  AdC7-HIVgp140 should be stored at ≤ -65°C prior to use/preparation.
  The study product is described in further detail in the IB.
  Arms: Part A, Group 2: AdC7-HIVgp140; Part B, Group 4: AdC6-HIVgp140 + AdC7-HIVgp140 + 400 mcg CH505TF gp120/GLA-SE; Part B, Group 5: AdC7-HIVgp140 + AdC6-HIVgp140 + 400 mcg CH505TF gp120/GLA-SE
Biological: CH505TF gp120 — CH505TF gp120 is formulated in 20 mM sodium phosphate, 150 mM NaCl, 0.02% polysorbate 80 (PS80), pH 6.5, supplied as a frozen liquid in 2 mL glass vials. Each 2 mL vial contains 0.75 mL of formulated gp120 at a concentration of 0.8 mg/mL and is stored at ≤ -65°C.
  The study product is described in further detail in the IB.
  Arms: Part B, Group 4: AdC6-HIVgp140 + AdC7-HIVgp140 + 400 mcg CH505TF gp120/GLA-SE; Part B, Group 5: AdC7-HIVgp140 + AdC6-HIVgp140 + 400 mcg CH505TF gp120/GLA-SE
Biological: GLA-SE (glucopyranosyl lipid A - stable emulsion; [labeled as AP 10-201]) — The GLA-SE adjuvant will be provided as vials containing 20 mcg/mL GLA in a 4% oil-in-water emulsion. Each sterile, single use vial contains 0.4 mL of product. Product appears as a milky-white liquid. GLA-SE must be stored at 2° to 8°C and must not be frozen. The study product is described in further detail within the IB.
  Arms: Part B, Group 4: AdC6-HIVgp140 + AdC7-HIVgp140 + 400 mcg CH505TF gp120/GLA-SE; Part B, Group 5: AdC7-HIVgp140 + AdC6-HIVgp140 + 400 mcg CH505TF gp120/GLA-SE
Biological: Placebo — Placebo will be Sodium Chloride for Injection, 0.9%, will be used as the placebo. It must be stored as recommended by the manufacturer.
  Arms: Part A, Group 3: Placebo; Part B, Group 6: Placebo + Placebo + Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of HIV-1 vaccines based on chimpanzee serotypes of adenovirus expressing clade C gp140 and a CH505TF gp120 protein boost in healthy, HIV- uninfected adult participants.

DETAILED DESCRIPTION:
This study will evaluate the safety and tolerability of AdC6-HIVgp140 and AdC7-HIVgp140 at doses of 1 x 10^10 virus particles (vp) and 5 x 10^10 vp, alone and in combination with CH505TF gp120 adjuvanted with GLA-SE in HIV- uninfected adults.

Participants will be randomly assigned to 6 groups, separated into low dose (Part A; Groups 1-3) and high dose (Part B; Groups 4-6).

Participants in Group 1 (Groups 1-3) will receive 1 x 10^10 vp of AdC6-HIVgp140. Participants in Group 2 will receive 1 x 10^10 vp of AdC7-HIVgp140. Participants in Group 3 will receive Placebo control.

Part A participants will undergo 6 months of scheduled clinic visits (main study) followed by AESI (Adverse Events of Special Interest) health contacts at month 12, and then annual health contacts at month 24 and 36.

Participants in Group 4 will receive 5 x 10^10 vp of AdC6-HIVgp140 followed by 5 x 10^10 vp of AdC7-HIVgp140 (month 3) and 400 mcg CH505TF with 10 mcg GLA-SE (month 6). Participants in Group 5 will receive 5 x 10^10 vp of AdC7-HIVgp140 followed by 5 x 10^10 vp of AdC6-HIVgp140 (month 3) and 400 mcg CH505TF with 10 mcg GLA-SE (month 6). Participants in Group 6 will receive Placebo control.

Part B participants (Group 4-6) will undergo 12 months of scheduled clinic visits (main study) followed by an AESI health contact at month 18, and then annual health contacts at month 24 and 36.

ELIGIBILITY:
Inclusion Criteria:

General and Demographic Criteria

* Age of 18 through 50 years.
* Access to a participating HVTN CRS and willingness to be followed for the planned duration of the study.
* Ability and willingness to provide informed consent.
* Assessment of understanding: volunteer demonstrates understanding of this study and that in a previous trial with an adenovirus type 5 (Ad5) vector there was an association of increased HIV acquisition with receipt of that study product; completes a questionnaire prior to first vaccination with verbal demonstration of understanding of all questionnaire items answered incorrectly.
* Willing to be contacted annually after completion of scheduled clinic visits for a total of 3 years following initial study injection.
* Agrees not to enroll in another study of an investigational research agent until the last scheduled clinic visit.
* Good general health as shown by medical history, physical exam, and screening laboratory tests.

HIV-Related Criteria

* Willingness to receive HIV test results.
* Willingness to discuss HIV infection risks and amenable to HIV risk reduction counseling.
* Assessed as "low risk" for HIV acquisition per low risk guidelines (see Appendix M), agrees to discuss HIV infection risks, agrees to risk reduction counseling, and agrees to avoid behavior associated with high risk of HIV exposure through the final study visit. Low risk may include persons stably taking PrEP as prescribed for 6 months or longer.

Laboratory Inclusion Values

Hemogram/Complete blood count (CBC)

* Hemoglobin

  * 11.0 g/dL for volunteers who were assigned female sex at birth
  * 13.0 g/dL for volunteers who were assigned male sex at birth and transgender male who have been on hormone therapy for more than 6 consecutive months
  * 12.0 g/dL for transgender female who have been on hormone therapy for more than 6 consecutive months

For transgender participants who have been on hormone therapy for less than 6 consecutive months, determine hemoglobin eligibility based on the sex assigned at birth

* White blood cell count = 2,500 to 12,000 cells/mm3 with normal differential, or differential approved by Investigator of Record (IoR) or designee as not clinically significant
* Total lymphocyte count ≥ 650 cells/mm3 with normal differential, or differential approved by Investigator of Record (IoR) or designee as not clinically significant
* Remaining differential either within institutional normal range or with site physician approval.
* Platelets = 125,000 to 550,000 cells/mm3.

Chemistry

* Alanine aminotransferase (ALT) < 1.25 times the institutional upper limit of normal;
* Creatinine <1.1 times the institutional upper limit of normal

Virology

* Negative HIV-1 and -2 blood test: US volunteers must have a negative FDA-approved enzyme immunoassay (EIA) or chemiluminescent microparticle immunoassay (CMIA).
* Negative Hepatitis B surface antigen (HBsAg).
* Negative anti-Hepatitis C virus antibodies (anti-HCV), or negative HCV nucleic acid test if the anti-HCV is positive

Urine

* Normal urine:

  * Negative or trace urine protein, and
  * Negative, trace, or 1+ blood/hemoglobin on urine dipstick. If 1+ hemoglobin is present on dipstick, a microscopic urinalysis with red blood cells levels within institutional normal range is required.

Reproductive Status

* Volunteers who were assigned female sex at birth: negative serum or urine beta human chorionic gonadotropin (β-HCG) pregnancy test at screening (ie, prior to randomization) and prior to study product administration on the day of study product administration. Persons who are NOT of reproductive potential due to having undergone hysterectomy or bilateral oophorectomy (verified by medical records), are not required to undergo pregnancy testing.
* Reproductive status: A volunteer who was assigned female sex at birth must agree to use effective contraception for sexual activity that could lead to pregnancy from at least 21 days prior to enrollment until two months following final product administration.

  * Condoms (male or female) with or without a spermicide,
  * Diaphragm or cervical cap with spermicide,
  * Intrauterine device (IUD),
  * Hormonal contraception,
  * Tubal ligation, or
  * Any other contraceptive method approved by the HVTN 139 PSRT
  * Successful vasectomy in any partner assigned male sex at birth (considered successful if a volunteer reports that a male partner has [1] documentation of azoospermia by microscopy, or [2] a vasectomy more than 2 years ago with no resultant pregnancy despite sexual activity postvasectomy);
  * Or not be of reproductive potential, such as having reached menopause (no menses for 1 year) or having undergone hysterectomy, or bilateral oophorectomy;
  * Or be sexually abstinent.
* Volunteers who were assigned female sex at birth must also agree not to seek pregnancy through alternative methods, such as artificial insemination or in vitro fertilization until two months after the last product administration

Exclusion Criteria:

* Blood products received within 120 days before first vaccination.
* Investigational research agents received within 30 days before first vaccination.
* Body mass index (BMI) ≥ 40; or BMI ≥ 35 with 2 or more of the following: age > 45, systolic blood pressure > 140 mm Hg, diastolic blood pressure > 90 mm Hg, current tobacco smoker, known hyperlipidemia.
* Intent to participate in another study of an investigational research agent or any other study that requires non-HVTN HIV antibody testing during the planned duration of the HVTN 139 study.
* Pregnant or breastfeeding.
* Active duty and reserve US military personnel.

Vaccines and other Injections

* HIV vaccine(s) received in a prior HIV vaccine trial. For volunteers who have received control/placebo in an HIV vaccine trial, the HVTN 139 PSRT will determine eligibility on a case-by-case basis.
* Previous receipt of monoclonal antibodies (mAbs), whether licensed or investigational. Exceptions may be made by the HVTN 139 PSRT on a case-by-case basis.
* Non-HIV experimental vaccine(s) received within the last 1 year in a prior vaccine trial. Exceptions may be made by the HVTN 139 PSRT for vaccines that have subsequently undergone licensure by the FDA. For volunteers who have received control/placebo in an experimental vaccine trial, the HVTN 139 PSRT will determine eligibility on a case-by-case basis. For volunteers who have received an experimental vaccine(s) greater than 1 years ago, eligibility for enrollment will be determined by the HVTN 139 PSRT on a case-by-case basis.
* Live attenuated vaccines received within 30 days before first vaccination or scheduled within 28 days after injection (eg, measles, mumps, and rubella [MMR]; oral polio vaccine [OPV]; varicella; yellow fever; live attenuated influenza vaccine).
* Any vaccines that are not live attenuated vaccines and were received within 14 days prior to first vaccination (eg, tetanus, pneumococcal, Hepatitis A or B).
* Allergy treatment with antigen injections within 30 days before first vaccination or that are scheduled within 14 days after first vaccination.

Immune System

* Immunosuppressive medications received within 168 days before first vaccination (Not exclusionary: [1] corticosteroid nasal spray; [2] inhaled corticosteroids; [3] topical corticosteroids for mild, uncomplicated dermatologic condition; or [4] a single course of oral/parenteral prednisone or equivalent at doses < 60 mg/day and length of therapy < 11 days with completion at least 30 days prior to enrollment).
* Serious adverse reactions to vaccines or to vaccine components such as glycerol, sodium chloride, tris (hydroxymethyl)aminomethane including history of anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain. (Not excluded from participation: a volunteer who had a nonanaphylactic adverse reaction to pertussis vaccine as a child).
* Immunoglobulin received within 90 days before first vaccination (for mAb see criterion 8 above).
* Autoimmune disease, current or history. (Not exclusionary: well-controlled psoriasis that does not require systemic therapy)
* AESIs

Volunteers who currently have, or have a history of, any condition that could be considered an AESI for the products administered in this protocol (representative examples are listed in Appendix N). The exception to Appendix N is well-controlled psoriasis, which is not exclusionary (as above)

* Immunodeficiency.

Clinical significant medical conditions

* Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health. A clinically significant condition or process includes but is not limited to:

  * A process that would affect the immune response,
  * A process that would require medication that affects the immune response,
  * Any contraindication to repeated injections or blood draws,
  * A condition that requires active medical intervention or monitoring to avert grave danger to the volunteer's health or well-being during the study period,
  * A condition or process for which signs or symptoms could be confused with reactions to vaccine, or
  * Any condition specifically listed among the exclusion criteria below.
* Any medical, psychiatric, occupational, or other condition that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety or reactogenicity, or a volunteer's ability to give informed consent.
* Psychiatric condition that precludes compliance with the protocol. Specifically excluded are persons with psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years.
* Current anti-tuberculosis (TB) prophylaxis or therapy.
* Asthma exclusion criteria: Asthma is excluded if the participant has ANY of the following:

  * Required either oral or parenteral corticosteroids for an exacerbation two or more times within the past year; OR
  * Needed emergency care, urgent care, hospitalization, or intubation for asthma within the past year; OR
  * Uses a short-acting rescue inhaler more than 2 days/week; OR
  * Uses medium-to-high dose inhaled corticosteroids (greater than 250 mcg fluticasone or therapeutic equivalent) or more than one medication for maintenance therapy daily. For example, potential participants taking long acting bronchodilator/inhaled corticosteroid combinations for daily maintenance are excluded. [Note: Maintenance monotherapy with cromolyn, leukotriene receptor antagonist, or theophylline is not exclusionary.]; OR
  * Meets any other asthma-related criteria that, in the judgement of the investigator, could lead to interference with study participation.
* Diabetes mellitus type 1 or type 2. (Not exclusionary: type 2 cases controlled with diet alone or a history of isolated gestational diabetes)
* Thyroidectomy, or thyroid disease (Not exclusionary: well-controlled non-autoimmune thyroid disease as defined in HVTN 139 Study Specific Procedures (SSP))
* Hypertension:

If a person has been found to have elevated blood pressure or hypertension during screening or previously, exclude for blood pressure that is not well controlled. Well-controlled blood pressure is defined in this protocol as consistently < 140 mm Hg systolic and < 90 mm Hg diastolic, with or without medication, with only isolated, brief instances of higher readings, which must be ≤ 150 mm Hg systolic and ≤ 100 mm Hg diastolic. For these volunteers, blood pressure must be < 140 mm Hg systolic and < 90 mm Hg diastolic at enrollment.

If a person has NOT been found to have elevated blood pressure or hypertension during screening or previously, exclude for systolic blood pressure ≥ 150 mm Hg at enrollment or diastolic blood pressure ≥ 100 mm Hg at enrollment.

* Bleeding disorder (eg, factor deficiency, coagulopathy, or platelet disorder requiring special precautions)
* Malignancy (Not excluded from participation: Volunteer who has had malignancy excised surgically and who, in the investigator's estimation, has a reasonable assurance of sustained cure, or who is unlikely to experience recurrence of malignancy during the period of the study).
* Seizure disorder: History of seizure(s) within past three years. Also exclude if volunteer has used medications in order to prevent or treat seizure(s) at any time within the past 3 years.
* Asplenia: any condition resulting in the absence of a functional spleen.
* History of angioedema, or anaphylaxis. (Not exclusionary: angioedema or anaphylaxis with known trigger and no episodes within five years.)
* History of generalized urticaria within past five years.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2021-11-25 (Actual); Primary Completion 2023-08-21 (Actual); Study Completion 2025-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ameena Goga, Study Chair — HIV Prevention Research Unit, South African Medical Research Council
Locations (6):
- South Africa (6):
  - Emavundleni CRS, Cape Town
  - CAPRISA eThekwini CRS, Durban
  - Isipingo CRS, Isipingo
  - Soweto HVTN CRS, Johannesburg
  - Aurum Institute Klerksdorp CRS, Klerksdorp
  - Setshaba Research Centre CRS, Soshanguve

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A, Group 1: Vaccine: AdC6-HIVgp140 1 x 10^10 vp to be administrated IM at Month 0
- Part A, Group 2: Vaccine: AdC7-HIVgp140 1 x 10^10 vp to be administrated IM at Month 0
- Part A, Group 3: Placebo: Placebo
  Control for AdC6-HIVgp140 or AdC7-HIVgp140, Sodium Chloride for Injection, 0.9%. Control for CH505TF gp120/GLA-SE adjuvanted protein: Sodium Chloride for Injection, 0.9%.
- Part B, Group 4: Vaccine: AdC6-HIVgp140 5 x 10^10 vp at Month 0 and AdC7-HIVgp140 5 x 10^10 vp at Month 3 and CH505TF/GLA-SE 400mg at Month 6
- Part B, Group 5: Vaccine: AdC7-HIVgp140 5 x 10^10 vp at Month 0 and AdC6-HIVgp140 5 x 10^10 vp at Month 3 and CH505TF/GLA-SE 400mg at Month 6
- Part B, Group 6: Placebo: Placebo+Placebo+Placebo
  Control for AdC6-HIVgp140 or AdC7-HIVgp140, Sodium Chloride for Injection, 0.9%. Control for CH505TF gp120/GLA-SE adjuvanted protein: Sodium Chloride for Injection, 0.9%.
Period: Overall Study
Arm/Group | Part A, Group 1: Vaccine | Part A, Group 2: Vaccine | Part A, Group 3: Placebo | Part B, Group 4: Vaccine | Part B, Group 5: Vaccine | Part B, Group 6: Placebo
Started ([1]Enrolled) | 5 | 5 | 2 | 10 | 10 | 2
Completed (Term form with reason = scheduled exit visit) | 5 | 5 | 2 | 9 | 7 | 2
Not Completed | 0 | 0 | 0 | 1 | 3 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Participant unable to adhere Visit Schedule | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A, Group 1: Vaccine | Part A, Group 2: Vaccine | Part A, Group 3: Placebo | Part B, Group 4: Vaccine | Part B, Group 5: Vaccine | Part B, Group 6: Placebo | Total
Number analyzed (Participants) | 5 | 5 | 2 | 10 | 10 | 2 | 34
Age, Continuous [Median (Full Range); unit: years] | 23 [19 to 36] | 23 [18 to 32] | 24.5 [21 to 28] | 28 [19 to 35] | 28 [18 to 40] | 21.5 [20 to 23] | 25.5 [18 to 40]
Age, Customized [Count of Participants; unit: Participants]
  Less than 18 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  18-20 | 2 | 2 | 0 | 1 | 1 | 1 | 7
  21-30 | 2 | 2 | 2 | 6 | 5 | 1 | 18
  31-40 | 1 | 1 | 0 | 3 | 4 | 0 | 9
  41-50 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Age Category : Above 50 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 0 | 3 | 5 | 0 | 12
  Male | 3 | 3 | 2 | 7 | 5 | 2 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 5 | 2 | 10 | 10 | 2 | 34
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 5 | 2 | 10 | 10 | 2 | 34
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 5 | 5 | 2 | 10 | 10 | 2 | 34
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Indian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Colored | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  South Africa | 5 | 5 | 2 | 10 | 10 | 2 | 34

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Local Reactogenicity Events Signs and Symptoms: Pain and/or Tenderness
Description: Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1 [July 2017]. The maximum grade observed for each symptom over the time frame is presented.
Time Frame: Measured through 7 days after each study product administration at Study Day 0 (Month 0) for Part A (T1, T2, and C3) and at Study Days 0 (Month 0), 84 (Month 3) and 168 (Month 6) for Part B (T4, T5, and C6).
Measure: Count of Participants; unit: Participants
Groups:
- Part A, Group 2: Vaccine: AdC7-HIVgp140 1 x 10^10 vp to be administrated IM at Month
Arm/Group | Part A, Group 1: Vaccine | Part A, Group 2: Vaccine | Part A, Group 3: Placebo | Part B, Group 4: Vaccine | Part B, Group 5: Vaccine | Part B, Group 6: Placebo
Number analyzed (Participants) | 5 | 5 | 2 | 10 | 10 | 2
Participants
  None | 5 | 4 | 1 | 6 | 5 | 2
  Mild | 0 | 1 | 1 | 4 | 2 | 0
  Moderate | 0 | 0 | 0 | 0 | 3 | 0
  Severe | 0 | 0 | 0 | 0 | 0 | 0
  Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants Reporting Local Reactogenicity Signs and Symptoms: Erythema and/or Induration
Description: as for outcome 1
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: Vaccine | Part A, Group 2: Vaccine | Part A, Group 3: Placebo | Part B, Group 4: Vaccine | Part B, Group 5: Vaccine | Part B, Group 6: Placebo
Number analyzed (Participants) | 5 | 5 | 2 | 10 | 10 | 2
Participants
  Erythema/Redness: None | 5 | 5 | 2 | 10 | 8 | 2
  Erythema/Redness: Mild | 0 | 0 | 0 | 0 | 2 | 0
  Erythema/Redness: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Erythema/Redness: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Erythema/Redness: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0
  Induration/Swelling: None | 5 | 5 | 2 | 10 | 10 | 2
  Induration/Swelling: Mild | 0 | 0 | 0 | 0 | 0 | 0
  Induration/Swelling: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Induration/Swelling: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Induration/Swelling: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants Reporting Systemic Reactogenicity Signs and Symptoms
Description: as for outcome 1
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: Vaccine | Part A, Group 2: Vaccine | Part A, Group 3: Placebo | Part B, Group 4: Vaccine | Part B, Group 5: Vaccine | Part B, Group 6: Placebo
Number analyzed (Participants) | 5 | 5 | 2 | 10 | 10 | 2
Participants
  Malaise and/or fatigue: None | 5 | 5 | 2 | 6 | 7 | 1
  Malaise and/or fatigue: Mild | 0 | 0 | 0 | 3 | 2 | 1
  Malaise and/or fatigue: Moderate | 0 | 0 | 0 | 1 | 1 | 0
  Malaise and/or fatigue: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Malaise and/or fatigue: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0
  Myalgia: None | 5 | 5 | 2 | 7 | 7 | 2
  Myalgia: Mild | 0 | 0 | 0 | 2 | 2 | 0
  Myalgia: Moderate | 0 | 0 | 0 | 1 | 1 | 0
  Myalgia: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Myalgia: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0
  Headache: None | 5 | 3 | 2 | 7 | 5 | 2
  Headache: Mild | 0 | 2 | 0 | 3 | 3 | 0
  Headache: Moderate | 0 | 0 | 0 | 0 | 2 | 0
  Headache: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Headache: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0
  Nausea: None | 5 | 5 | 2 | 7 | 9 | 2
  Nausea: Mild | 0 | 0 | 0 | 2 | 0 | 0
  Nausea: Moderate | 0 | 0 | 0 | 1 | 1 | 0
  Nausea: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Nausea: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0
  Chills: None | 5 | 4 | 2 | 9 | 6 | 2
  Chills: Mild | 0 | 1 | 0 | 0 | 3 | 0
  Chills: Moderate | 0 | 0 | 0 | 1 | 1 | 0
  Chills: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Chills: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0
  Arthralgia: None | 5 | 4 | 2 | 8 | 8 | 2
  Arthralgia: Mild | 0 | 1 | 0 | 1 | 0 | 0
  Arthralgia: Moderate | 0 | 0 | 0 | 1 | 2 | 0
  Arthralgia: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Arthralgia: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0
  Temperature: None | 5 | 5 | 2 | 10 | 8 | 2
  Temperature: Mild | 0 | 0 | 0 | 0 | 2 | 0
  Temperature: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Temperature: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Temperature: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0
  Max. Systemic Symptoms: None | 5 | 3 | 2 | 5 | 4 | 1
  Max. Systemic Symptoms: Mild | 0 | 2 | 0 | 4 | 3 | 1
  Max. Systemic Symptoms: Moderate | 0 | 0 | 0 | 1 | 3 | 0
  Max. Systemic Symptoms: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Max. Systemic Symptoms: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Numbers of Participant With Early Study Termination Associated With Reactogenicity, AE, or Death During Main Study and AESI Visits.
Description: From the termination and adverse event forms that were collected during main study clinical visits period and AESI contact visits. Counts are tabulated by treatment arm.
Time Frame: Early study termination reason was collected through 7 days for reactogenicity, 30 days for AEs and 12 months for deaths following any receipt of study product (up to 18 months).
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: Vaccine | Part A, Group 2: Vaccine | Part A, Group 3: Placebo | Part B, Group 4: Vaccine | Part B, Group 5: Vaccine | Part B, Group 6: Placebo
Number analyzed (Participants) | 5 | 5 | 2 | 10 | 10 | 2
Participants | 0 | 0 | 0 | 0 | 1 | 0

5. Primary Outcome: Number of Participants Reporting Serious Adverse Events (SAEs)
Description: From adverse event (AE) forms, counts are tabulated by treatment arm. AE forms were collected during main study clinical visits and AESI contact visits
Time Frame: Measured through 12 months following any receipt of study product(up to 18 months). Study products were given at Study Day 0 (Month 0) for Part A (T1, T2, and C3) and at Study Days 0 (Month 0), 84 (Month 3) and 168 (Month 6) for Part B (T4, T5, and C6).
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: Vaccine | Part A, Group 2: Vaccine | Part A, Group 3: Placebo | Part B, Group 4: Vaccine | Part B, Group 5: Vaccine | Part B, Group 6: Placebo
Number analyzed (Participants) | 5 | 5 | 2 | 10 | 10 | 2
Participants | 0 | 0 | 0 | 0 | 1 | 0

6. Primary Outcome: Number of Participants Reporting Medically Attended Adverse Events (MAAEs)
Description: as for outcome 5
Time Frame: as for outcome 5
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: Vaccine | Part A, Group 2: Vaccine | Part A, Group 3: Placebo | Part B, Group 4: Vaccine | Part B, Group 5: Vaccine | Part B, Group 6: Placebo
Number analyzed (Participants) | 5 | 5 | 2 | 10 | 10 | 2
Participants | 0 | 1 | 0 | 1 | 0 | 0

7. Primary Outcome: Number of Participants Reporting Adverse Event of Special Interests (AESIs)
Description: as for outcome 5
Time Frame: as for outcome 5
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: Vaccine | Part A, Group 2: Vaccine | Part A, Group 3: Placebo | Part B, Group 4: Vaccine | Part B, Group 5: Vaccine | Part B, Group 6: Placebo
Number analyzed (Participants) | 5 | 5 | 2 | 10 | 10 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Response Rate of HIV-specific Serum IgG Binding Antibodies Assessed 4 Weeks After a Single Vaccination (Part A) or the First Vaccination (Part B)
Description: Serum HIV-1-specific IgG responses (dilution 1:50) against gp120, gp140, gp70-V1V2 and gp41 antigens were measured on a Bio-Plex instrument (Bio-Rad) using a standardized custom HIV-1 Luminex assay. The readout was background-subtracted mean fluorescence intensity (MFI), where background referred to a plate level control (i.e., a blank well run on each plate). Samples from post-enrollment visits were declared to have positive responses if they met three conditions: (1) the mean fluorescence intensity (MFI) minus blank (MFI*) values were ≥ antigen-specific cutoff at the 1:50 dilution level (based on the 95th percentile of baseline samples as calculated by SAS PROC UNIVARIATE default method, and at least 100 MFI minus blank), (2) the MFI minus blank values were greater than 3 times the baseline (day 0) MFI minus blank values, and (3) the MFI values were greater than 3 times the baseline MFI values.
Time Frame: Measured at Month 1 for both Part A and Part B
Population: Overall Number of Participants Analyzed represents the number participants with specimen at Month 1. Number Analyzed-shows the number of participants with available data after filtering for assay specific quality control criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: Vaccine | Part A, Group 2: Vaccine | Part A, Group 3: Placebo | Part B, Group 4: Vaccine | Part B, Group 5: Vaccine | Part B, Group 6: Placebo
Number analyzed (Participants) | 4 | 4 | 2 | 10 | 8 | 2
Participants
  1086C_D7gp120.avi/293F measured at Month 1 | 4 | 2 | 0 | 6 | 5 | 0
  1394C9_G1.D11gp120.avi measured at Month 1 | 0 | 0 | 0 | 0 | 0 | 0
  1428_D11gp120.avi/293F measured at Month 1: number analyzed (Participants) | 4 | 4 | 2 | 10 | 7 | 2
  1428_D11gp120.avi/293F measured at Month 1 | 0 | 0 | 0 | 1 | 0 | 0
  1641A7_D11gp120.avi/293F measured at Month 1 | 0 | 0 | 0 | 3 | 1 | 0
  96ZM651.D11gp120.avi measured at Month 1: number analyzed (Participants) | 4 | 4 | 2 | 10 | 7 | 1
  96ZM651.D11gp120.avi measured at Month 1 | 0 | 0 | 0 | 0 | 0 | 0
  CAP210_D11gp120.avi/293F measured at Month 1: number analyzed (Participants) | 4 | 4 | 2 | 10 | 7 | 2
  CAP210_D11gp120.avi/293F measured at Month 1 | 0 | 0 | 0 | 1 | 0 | 0
  CAP45_D11gp120.avi/293F measured at Month 1 | 0 | 0 | 0 | 1 | 0 | 0
  CH0505_CON D7gp120_avi/293F/Mon measured at Month 1: number analyzed (Participants) | 4 | 4 | 2 | 10 | 7 | 2
  CH0505_CON D7gp120_avi/293F/Mon measured at Month 1 | 0 | 0 | 0 | 0 | 0 | 0
  CH505TF D7gp120d371_avi/293F/Mon measured at Month 1: number analyzed (Participants) | 4 | 4 | 2 | 10 | 7 | 2
  CH505TF D7gp120d371_avi/293F/Mon measured at Month 1 | 0 | 0 | 0 | 0 | 0 | 0
  CH505TFD8N156KN160K_avi/293i Mon measured at Month 1: number analyzed (Participants) | 4 | 4 | 2 | 10 | 7 | 1
  CH505TFD8N156KN160K_avi/293i Mon measured at Month 1 | 0 | 0 | 0 | 1 | 0 | 0
  Ce0042_D11gp120.avi/293F measured at Month 1: number analyzed (Participants) | 4 | 4 | 2 | 10 | 7 | 2
  Ce0042_D11gp120.avi/293F measured at Month 1 | 0 | 0 | 0 | 0 | 0 | 0
  Con 6 gp120/B measured at Month 1 | 0 | 1 | 0 | 1 | 2 | 0
  Con S gp140 CFI measured at Month 1 | 1 | 1 | 0 | 9 | 3 | 0
  Du156_D11gp120.avi/293F measured at Month 1 | 1 | 0 | 0 | 7 | 2 | 0
  TV1c8_D11gp120.avi/293F measured at Month 1 | 1 | 0 | 0 | 8 | 2 | 0
  gp41 measured at Month 1: number analyzed (Participants) | 4 | 3 | 2 | 10 | 6 | 2
  gp41 measured at Month 1 | 2 | 0 | 0 | 8 | 3 | 0
  gp70-001428.2.42 V1V2 measured at Month 1: number analyzed (Participants) | 4 | 4 | 2 | 9 | 7 | 2
  gp70-001428.2.42 V1V2 measured at Month 1 | 0 | 0 | 0 | 0 | 2 | 0
  gp70-1012.11.TC21.3257 V1V2 measured at Month 1: number analyzed (Participants) | 4 | 4 | 2 | 9 | 6 | 2
  gp70-1012.11.TC21.3257 V1V2 measured at Month 1 | 0 | 0 | 0 | 0 | 2 | 0
  gp70-1051.12.C22 V1V2 measured at Month 1: number analyzed (Participants) | 4 | 4 | 2 | 9 | 6 | 2
  gp70-1051.12.C22 V1V2 measured at Month 1 | 0 | 0 | 0 | 0 | 2 | 0
  gp70-1394C9G1 V1V2 measured at Month 1: number analyzed (Participants) | 4 | 4 | 2 | 9 | 7 | 2
  gp70-1394C9G1 V1V2 measured at Month 1 | 0 | 0 | 0 | 0 | 2 | 0
  gp70-7060101641 V1V2 measured at Month 1: number analyzed (Participants) | 4 | 4 | 2 | 9 | 7 | 2
  gp70-7060101641 V1V2 measured at Month 1 | 0 | 0 | 0 | 0 | 0 | 0
  gp70-96ZM651.02 V1v2 measured at Month 1: number analyzed (Participants) | 4 | 4 | 2 | 9 | 7 | 2
  gp70-96ZM651.02 V1v2 measured at Month 1 | 1 | 0 | 0 | 4 | 1 | 0
  gp70-BF1266_431a_V1V2 measured at Month 1: number analyzed (Participants) | 4 | 4 | 2 | 9 | 6 | 2
  gp70-BF1266_431a_V1V2 measured at Month 1 | 0 | 0 | 0 | 0 | 2 | 0
  gp70-CAP210.2.00.E8 V1V2 measured at Month 1: number analyzed (Participants) | 4 | 4 | 2 | 9 | 7 | 2
  gp70-CAP210.2.00.E8 V1V2 measured at Month 1 | 0 | 1 | 0 | 0 | 3 | 0
  gp70-CAP45.2.00.G3 V1V2 measured at Month 1: number analyzed (Participants) | 4 | 4 | 2 | 9 | 7 | 2
  gp70-CAP45.2.00.G3 V1V2 measured at Month 1 | 0 | 0 | 0 | 0 | 1 | 0
  gp70-Ce1086_B2 V1V2 measured at Month 1: number analyzed (Participants) | 4 | 4 | 2 | 9 | 7 | 2
  gp70-Ce1086_B2 V1V2 measured at Month 1 | 0 | 0 | 0 | 1 | 1 | 0
  gp70-Ce1176 V1V2 measured at Month 1: number analyzed (Participants) | 4 | 4 | 2 | 9 | 7 | 2
  gp70-Ce1176 V1V2 measured at Month 1 | 0 | 1 | 0 | 0 | 2 | 0
  gp70-Ce704010042_2ES V1V2 measured at Month 1: number analyzed (Participants) | 4 | 4 | 2 | 9 | 7 | 2
  gp70-Ce704010042_2ES V1V2 measured at Month 1 | 0 | 0 | 0 | 0 | 0 | 0
  gp70-ConC V1V2 measured at Month 1: number analyzed (Participants) | 4 | 4 | 2 | 9 | 7 | 2
  gp70-ConC V1V2 measured at Month 1 | 0 | 0 | 0 | 0 | 1 | 0
  gp70-Du156.12 V1V2 measured at Month 1: number analyzed (Participants) | 4 | 4 | 2 | 9 | 7 | 2
  gp70-Du156.12 V1V2 measured at Month 1 | 0 | 0 | 0 | 0 | 0 | 0
  gp70-TV1.21 V1V2 measured at Month 1: number analyzed (Participants) | 4 | 4 | 2 | 9 | 6 | 2
  gp70-TV1.21 V1V2 measured at Month 1 | 1 | 1 | 0 | 0 | 2 | 0
  gp70_CH505TF_V1V2_N156KN160K_avi/293F measured at Month 1: number analyzed (Participants) | 4 | 4 | 2 | 9 | 6 | 1
  gp70_CH505TF_V1V2_N156KN160K_avi/293F measured at Month 1 | 0 | 0 | 0 | 0 | 0 | 0
  gp70_CH505TF_V1V2_avi/293F measured at Month 1: number analyzed (Participants) | 3 | 3 | 2 | 9 | 6 | 1
  gp70_CH505TF_V1V2_avi/293F measured at Month 1 | 0 | 0 | 0 | 0 | 1 | 0

9. Secondary Outcome: Magnitude of HIV-specific Serum IgG Binding Antibodies Assessed 4 Weeks After a Single Vaccination (Part A) or the First Vaccination (Part B)
Description: Serum HIV-1-specific IgG responses (dilution 1:50) against gp120, gp140, gp70-V1V2 and gp41 antigens were measured on a Bio-Plex instrument (Bio-Rad) using a standardized custom HIV-1 Luminex assay. The readout was background-subtracted mean fluorescence intensity (MFI), where background referred to a plate level control (i.e., a blank well run on each plate).
Time Frame: Measured at Month 1 for both Part A and Part B
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: Net MFI
Arm/Group | Part A, Group 1: Vaccine | Part A, Group 2: Vaccine | Part A, Group 3: Placebo | Part B, Group 4: Vaccine | Part B, Group 5: Vaccine | Part B, Group 6: Placebo
Number analyzed (Participants) | 4 | 4 | 2 | 10 | 8 | 2
Net MFI
  1086C_D7gp120.avi/293F measured at Month 1 | 691.2 [435 to 907.1] | 65.8 [7.4 to 229.6] | 1 [1 to 1] | 371.8 [153.4 to 1041.7] | 164.5 [1 to 612.6] | 8.1 [4.6 to 11.7]
  1394C9_G1.D11gp120.avi measured at Month 1 | 3.5 [1 to 27.1] | 1.2 [1 to 2.6] | 1 [1 to 1] | 22.2 [3.2 to 35.6] | 40.9 [1 to 144.7] | 1 [1 to 1]
  1428_D11gp120.avi/293F measured at Month 1: number analyzed (Participants) | 4 | 4 | 2 | 10 | 7 | 2
  1428_D11gp120.avi/293F measured at Month 1 | 1 [1 to 165.8] | 57.4 [16.4 to 341.9] | 1 [1 to 1] | 178.6 [122.2 to 539.3] | 3 [1 to 210.1] | 1874 [937.5 to 2810.5]
  1641A7_D11gp120.avi/293F measured at Month 1 | 1 [1 to 87.8] | 25.1 [1 to 52.8] | 1 [1 to 1] | 238.6 [116.8 to 921.8] | 23 [1 to 402.4] | 92.5 [46.8 to 138.2]
  96ZM651.D11gp120.avi measured at Month 1: number analyzed (Participants) | 4 | 4 | 2 | 10 | 7 | 1
  96ZM651.D11gp120.avi measured at Month 1 | 54.8 [36.2 to 724.5] | 186.9 [82 to 2016.1] | 1 [1 to 1] | 497.1 [89.9 to 851.5] | 27 [1 to 884.4] | 1 [1 to 1]
  CAP210_D11gp120.avi/293F measured at Month 1: number analyzed (Participants) | 4 | 4 | 2 | 10 | 7 | 2
  CAP210_D11gp120.avi/293F measured at Month 1 | 68.6 [1 to 317.6] | 81.9 [32.7 to 438.2] | 1 [1 to 1] | 291.5 [58.6 to 469.1] | 1 [1 to 458.9] | 2725.2 [1363.1 to 4087.4]
  CAP45_D11gp120.avi/293F measured at Month 1 | 25.4 [11.9 to 80.1] | 7.1 [2.1 to 51.2] | 1 [1 to 1] | 89.6 [61.2 to 280.8] | 41.8 [1 to 101.6] | 345.8 [173.4 to 518.1]
  CH0505_CON D7gp120_avi/293F/Mon measured at Month 1: number analyzed (Participants) | 4 | 4 | 2 | 10 | 7 | 2
  CH0505_CON D7gp120_avi/293F/Mon measured at Month 1 | 71.6 [1 to 281.5] | 336.5 [16.6 to 801.2] | 1 [1 to 1] | 137 [1 to 230] | 1 [1 to 131.9] | 3306.9 [1653.9 to 4959.8]
  CH505TF D7gp120d371_avi/293F/Mon measured at Month 1: number analyzed (Participants) | 4 | 4 | 2 | 10 | 7 | 2
  CH505TF D7gp120d371_avi/293F/Mon measured at Month 1 | 63.2 [1 to 248.2] | 347 [3.6 to 830.3] | 1 [1 to 1] | 136.1 [1 to 268.7] | 1 [1 to 60.6] | 3192 [1596.5 to 4787.5]
  CH505TFD8N156KN160K_avi/293i Mon measured at Month 1: number analyzed (Participants) | 4 | 4 | 2 | 10 | 7 | 1
  CH505TFD8N156KN160K_avi/293i Mon measured at Month 1 | 104.8 [1 to 348.7] | 292.6 [20.9 to 745.1] | 1 [1 to 1] | 124.5 [2.1 to 225.5] | 1 [1 to 206.4] | 1 [1 to 1]
  Ce0042_D11gp120.avi/293F measured at Month 1: number analyzed (Participants) | 4 | 4 | 2 | 10 | 7 | 2
  Ce0042_D11gp120.avi/293F measured at Month 1 | 103.2 [58.3 to 205.7] | 103 [95 to 273.9] | 23.9 [12.4 to 35.3] | 167.2 [113.2 to 208.2] | 109.2 [13.8 to 229.9] | 365.6 [183.3 to 547.9]
  Con 6 gp120/B measured at Month 1 | 38.9 [1 to 88.1] | 36.1 [4.9 to 91.8] | 1 [1 to 1] | 36.5 [8.2 to 45.3] | 1 [1 to 59.7] | 12 [6.5 to 17.5]
  Con S gp140 CFI measured at Month 1 | 436.5 [255.8 to 1292.8] | 272.1 [23.4 to 645.4] | 8.6 [4.8 to 12.4] | 3530.2 [1597.1 to 13418.8] | 650.2 [242.9 to 3709] | 575 [312.2 to 837.8]
  Du156_D11gp120.avi/293F measured at Month 1 | 61.9 [44.1 to 806.5] | 7.9 [1 to 16.2] | 1 [1 to 1] | 615.2 [418.6 to 1879.2] | 14 [1 to 383.9] | 62 [31.5 to 92.5]
  TV1c8_D11gp120.avi/293F measured at Month 1 | 101.9 [11.5 to 1434] | 1 [1 to 26.8] | 1 [1 to 1] | 1227.5 [650.2 to 3362.1] | 20.6 [1 to 199.2] | 152 [76.5 to 227.5]
  gp41 measured at Month 1: number analyzed (Participants) | 4 | 3 | 2 | 10 | 6 | 2
  gp41 measured at Month 1 | 5349.6 [3079.3 to 11108.9] | 3582.8 [3573.8 to 3855.2] | 2214.9 [1902.8 to 2526.9] | 22000 [9936.3 to 22000] | 13128 [6580.5 to 16682.2] | 1268.5 [882.1 to 1654.9]
  gp70-001428.2.42 V1V2 measured at Month 1: number analyzed (Participants) | 4 | 4 | 2 | 9 | 7 | 2
  gp70-001428.2.42 V1V2 measured at Month 1 | 1 [1 to 1] | 1 [1 to 17.9] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1149.1] | 1 [1 to 1]
  gp70-1012.11.TC21.3257 V1V2 measured at Month 1: number analyzed (Participants) | 4 | 4 | 2 | 9 | 6 | 2
  gp70-1012.11.TC21.3257 V1V2 measured at Month 1 | 1 [1 to 230.9] | 1 [1 to 22.2] | 1 [1 to 1] | 1 [1 to 1] | 79 [1 to 238.4] | 1 [1 to 1]
  gp70-1051.12.C22 V1V2 measured at Month 1: number analyzed (Participants) | 4 | 4 | 2 | 9 | 6 | 2
  gp70-1051.12.C22 V1V2 measured at Month 1 | 1 [1 to 1] | 1 [1 to 42.9] | 1 [1 to 1] | 1 [1 to 1] | 41.6 [1 to 304.6] | 1 [1 to 1]
  gp70-1394C9G1 V1V2 measured at Month 1: number analyzed (Participants) | 4 | 4 | 2 | 9 | 7 | 2
  gp70-1394C9G1 V1V2 measured at Month 1 | 1 [1 to 1] | 1 [1 to 54.9] | 22.9 [11.9 to 33.8] | 1 [1 to 1] | 1 [1 to 692.1] | 1 [1 to 1]
  gp70-7060101641 V1V2 measured at Month 1: number analyzed (Participants) | 4 | 4 | 2 | 9 | 7 | 2
  gp70-7060101641 V1V2 measured at Month 1 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 251.2] | 1 [1 to 1]
  gp70-96ZM651.02 V1v2 measured at Month 1: number analyzed (Participants) | 4 | 4 | 2 | 9 | 7 | 2
  gp70-96ZM651.02 V1v2 measured at Month 1 | 443.5 [37.2 to 1604.8] | 2.5 [1 to 96.8] | 1 [1 to 1] | 679.8 [434.8 to 2164.2] | 365.2 [112.4 to 1161.6] | 1 [1 to 1]
  gp70-BF1266_431a_V1V2 measured at Month 1: number analyzed (Participants) | 4 | 4 | 2 | 9 | 6 | 2
  gp70-BF1266_431a_V1V2 measured at Month 1 | 26.8 [1 to 330.1] | 1.6 [1 to 78.2] | 1 [1 to 1] | 1 [1 to 1] | 166.5 [1 to 913.2] | 1 [1 to 1]
  gp70-CAP210.2.00.E8 V1V2 measured at Month 1: number analyzed (Participants) | 4 | 4 | 2 | 9 | 7 | 2
  gp70-CAP210.2.00.E8 V1V2 measured at Month 1 | 1 [1 to 35.4] | 65.2 [43.9 to 618.6] | 1 [1 to 1] | 1 [1 to 1] | 263.5 [66.2 to 965.2] | 1 [1 to 1]
  gp70-CAP45.2.00.G3 V1V2 measured at Month 1: number analyzed (Participants) | 4 | 4 | 2 | 9 | 7 | 2
  gp70-CAP45.2.00.G3 V1V2 measured at Month 1 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 636.2] | 1 [1 to 1]
  gp70-Ce1086_B2 V1V2 measured at Month 1: number analyzed (Participants) | 4 | 4 | 2 | 9 | 7 | 2
  gp70-Ce1086_B2 V1V2 measured at Month 1 | 29.9 [1 to 61.3] | 1 [1 to 251.9] | 1 [1 to 1] | 6.5 [1 to 81.5] | 1 [1 to 533] | 1 [1 to 1]
  gp70-Ce1176 V1V2 measured at Month 1: number analyzed (Participants) | 4 | 4 | 2 | 9 | 7 | 2
  gp70-Ce1176 V1V2 measured at Month 1 | 1 [1 to 1] | 70.2 [13 to 360.2] | 1 [1 to 1] | 1 [1 to 1] | 232.2 [12 to 452.5] | 1 [1 to 1]
  gp70-Ce704010042_2ES V1V2 measured at Month 1: number analyzed (Participants) | 4 | 4 | 2 | 9 | 7 | 2
  gp70-Ce704010042_2ES V1V2 measured at Month 1 | 1 [1 to 1] | 1 [1 to 7.2] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  gp70-ConC V1V2 measured at Month 1: number analyzed (Participants) | 4 | 4 | 2 | 9 | 7 | 2
  gp70-ConC V1V2 measured at Month 1 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 178.4] | 1 [1 to 1]
  gp70-Du156.12 V1V2 measured at Month 1: number analyzed (Participants) | 4 | 4 | 2 | 9 | 7 | 2
  gp70-Du156.12 V1V2 measured at Month 1 | 1 [1 to 1] | 1 [1 to 5.3] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  gp70-TV1.21 V1V2 measured at Month 1: number analyzed (Participants) | 4 | 4 | 2 | 9 | 6 | 2
  gp70-TV1.21 V1V2 measured at Month 1 | 1800.6 [1 to 3984.3] | 183.6 [37.2 to 1832.3] | 1 [1 to 1] | 1 [1 to 1] | 1173 [80.8 to 2925.8] | 15.8 [8.4 to 23.1]
  gp70_CH505TF_V1V2_N156KN160K_avi/293F measured at Month 1: number analyzed (Participants) | 4 | 4 | 2 | 9 | 6 | 1
  gp70_CH505TF_V1V2_N156KN160K_avi/293F measured at Month 1 | 425.9 [1 to 1156] | 59.6 [1 to 1378.8] | 1 [1 to 1] | 1 [1 to 13] | 62.2 [1 to 603.9] | 79.2 [79.2 to 79.2]
  gp70_CH505TF_V1V2_avi/293F measured at Month 1: number analyzed (Participants) | 3 | 3 | 2 | 9 | 6 | 1
  gp70_CH505TF_V1V2_avi/293F measured at Month 1 | 1 [1 to 2274.4] | 1 [1 to 150.6] | 1 [1 to 1] | 1 [1 to 322] | 929.6 [49.1 to 2142.9] | 283.2 [283.2 to 283.2]

10. Secondary Outcome: HIV-specific Serum IgG Binding Antibodies Magnitude Breadth of AUC (AUC--MB) by Panel and Treatment Arm Assessed 4 Weeks After a Single Vaccination (Part A) or the First Vaccination (Part B)
Description: The area under the magnitude-breadth curve (AUC-MB) was calculated by first measuring the mean fluorescence intensity (MFI) of antibody binding to each antigen at 1:50 dilution. For each sample, a magnitude-breadth curve is generated by plotting the number of antigens (breadth) that exceed a series of MFI thresholds (MFI >100). The area under this curve (AUC) is then computed by the trapezoidal rule to summarize both the strength and diversity of the antibody response in a single value, which is equivalent to the average of the log10 net MFI over the panel of antigens
Time Frame: Measured at Month 1 for both Part A and Part B
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: log10(net MFI)
Arm/Group | Part A, Group 1: Vaccine | Part A, Group 2: Vaccine | Part A, Group 3: Placebo | Part B, Group 4: Vaccine | Part B, Group 5: Vaccine | Part B, Group 6: Placebo
Number analyzed (Participants) | 4 | 4 | 2 | 10 | 8 | 2
log10(net MFI)
  Clade C gp120 measured at Month 1: number analyzed (Participants) | 4 | 4 | 2 | 10 | 7 | 1
  Clade C gp120 measured at Month 1 | 2 [2 to 2.08] | 2 [2 to 2] | 2 [2 to 2] | 2.19 [2.14 to 2.37] | 2 [2 to 2.09] | 2 [2 to 2]
  Clade C gp70 V1V2 measured at Month 1: number analyzed (Participants) | 4 | 4 | 2 | 9 | 6 | 2
  Clade C gp70 V1V2 measured at Month 1 | 2.05 [2 to 2.11] | 2 [2 to 2.07] | 2 [2 to 2] | 2 [2 to 2.12] | 2.12 [2.03 to 2.18] | 2 [2 to 2]

11. Secondary Outcome: Response Rate of HIV-specific CD4+ and CD8+ T-cell Responses Assessed 4 Weeks After a Single Vaccination (Part A) or the First Vaccination (Part B)
Description: The four entries in each table were the number of cells positive for IFN-γ and/or IL-2 for both the stimulated and the negative control data. If both negative control replicates were included, then the average number of total cells and the average number of positive cells were used. A one-sided Fisher's exact test was applied to the table, testing whether the number of cytokine-producing cells for the stimulated data was equal to that for the negative control data. Since multiple individual tests (for each peptide pool) were conducted simultaneously, a multiplicity adjustment was made to the two individual peptide pool p-values considered, using the Bonferroni-Holm adjustment method. If the adjusted p-value for a peptide pool was ≤ 0.00001, the response to the peptide pool for the T-cell subset was considered positive. If at least one peptide pool for a specific HIV-1 protein was positive, then the overall response to the protein was considered positive.
Time Frame: Measured at Month 1 for both Part A and Part B
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: Vaccine | Part A, Group 2: Vaccine | Part A, Group 3: Placebo | Part B, Group 4: Vaccine | Part B, Group 5: Vaccine | Part B, Group 6: Placebo
Number analyzed (Participants) | 4 | 4 | 2 | 9 | 8 | 2
Participants
  Any Env for CD4+ T Cells, measured at Month 1 | 1 | 3 | 0 | 3 | 7 | 0
  Any Env for CD8+ T Cells, measured at Month 1 | 1 | 2 | 1 | 5 | 5 | 0
  ENV-1-PTEG-SEQ for CD4+ T Cells, measured at Month 1 | 0 | 3 | 0 | 0 | 6 | 0
  ENV-1-PTEG-SEQ for CD8+ T Cells, measured at Month 1 | 1 | 2 | 1 | 4 | 4 | 0
  ENV-2-PTEG-SEQ for CD4+ T Cells, measured at Month 1 | 1 | 2 | 0 | 3 | 6 | 0
  ENV-2-PTEG-SEQ for CD8+ T Cells, measured at Month 1 | 0 | 1 | 0 | 1 | 4 | 0

12. Secondary Outcome: Magnitude of HIV-specific CD4+ and CD8+ T-cell by Cytokine, T-cell Subset, Antigen and Treatment Group Assessed 4 Weeks After a Single Vaccination (Part A) or the First Vaccination (Part B)
Description: PBMC samples were stimulated with synthetic peptide pools or left unstimulated as a negative control. For each sample, T-cell subset, and peptide pool, response magnitude is % cells expressing cytokines (IFNy and/or IL-2) after peptide stimulation minus % cells expressing markers after no stimulation. Reported responses magnitude for Any Env are the sum of ENV-1-PTEG-SEQ and ENV-2-PTEG-SEQ
Time Frame: Measured at Month 1 for both Part A and Part B
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: Percentage of cells
Arm/Group | Part A, Group 1: Vaccine | Part A, Group 2: Vaccine | Part A, Group 3: Placebo | Part B, Group 4: Vaccine | Part B, Group 5: Vaccine | Part B, Group 6: Placebo
Number analyzed (Participants) | 4 | 4 | 2 | 9 | 8 | 2
Percentage of cells
  Any Env for CD4+ T Cells, measured at Month 1 | 0.019 [0.005 to 0.043] | 0.103 [0.096 to 0.119] | 0.001 [0.001 to 0.001] | 0.028 [0.001 to 0.055] | 0.13 [0.053 to 0.162] | 0.011 [0.006 to 0.017]
  Any Env for CD8+ T Cells, measured at Month 1 | 0.011 [0.001 to 0.022] | 0.096 [0.035 to 0.189] | 0.028 [0.016 to 0.041] | 0.044 [0.007 to 0.091] | 0.067 [0.041 to 0.126] | 0.025 [0.021 to 0.029]
  ENV-1-PTEG-SEQ for CD4+ T Cells, measured at Month 1 | 0.008 [0.005 to 0.015] | 0.066 [0.047 to 0.084] | 0.001 [0.001 to 0.001] | 0.008 [0.001 to 0.019] | 0.047 [0.025 to 0.064] | 0.011 [0.006 to 0.016]
  ENV-1-PTEG-SEQ for CD8+ T Cells, measured at Month 1 | 0.011 [0.001 to 0.022] | 0.038 [0.025 to 0.11] | 0.017 [0.01 to 0.024] | 0.028 [0.007 to 0.033] | 0.033 [0.021 to 0.094] | 0.016 [0.009 to 0.022]
  ENV-2-PTEG-SEQ for CD4+ T Cells, measured at Month 1 | 0.011 [0.001 to 0.028] | 0.049 [0.037 to 0.058] | 0.001 [0.001 to 0.001] | 0.019 [0.001 to 0.036] | 0.065 [0.032 to 0.093] | 0.001 [0.001 to 0.001]
  ENV-2-PTEG-SEQ for CD8+ T Cells, measured at Month 1 | 0.001 [0.001 to 0.001] | 0.011 [0.007 to 0.035] | 0.012 [0.006 to 0.017] | 0.014 [0.001 to 0.023] | 0.023 [0.011 to 0.048] | 0.009 [0.006 to 0.012]

13. Secondary Outcome: Response Rate of Serum Neutralizing Antibodies Against Env-pseudotyped Vaccine Strains (Du422.1, Du172.17 and CH505TF) and a Tier 1A Neutralization Phenotype (MW965.26) Assessed 4 Weeks After a Single Vaccination (Part A) or the First Vaccination (Part B)
Description: Neutralizing antibodies against strains of HIV-1 were measured as a function of reductions in Tat-induced luciferase (Luc) reporter gene expression in TZMbl cells. A serum neutralization titer was defined as the serum dilution that reduced relative luminescence units (RLUs) by 50% and 80% (ID50 and ID80) relative to the RLUs in virus control wells (cells + virus only) after subtraction of background RLU (cells only). The assay performed in TZM-bl cells measured neutralization titers against the Env-pseudotyped vaccine strains (Du422.1, Du172.17 and CH505TF) and a virus that exhibits a tier 1A neutralization phenotype (MW965.26).
  Response to a virus/isolate was considered positive if the neutralization titer was at or above a pre-specified cutoff of 10.
Time Frame: Measured at Month 1 for both Part A and Part B
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: Vaccine | Part A, Group 2: Vaccine | Part A, Group 3: Placebo | Part B, Group 4: Vaccine | Part B, Group 5: Vaccine | Part B, Group 6: Placebo
Number analyzed (Participants) | 4 | 4 | 2 | 10 | 8 | 2
Participants
  CH505TF at dilution 50, measured at Month 1 | 0 | 1 | 0 | 1 | 0 | 0
  CH505TF at dilution 80, measured at Month 1 | 0 | 0 | 0 | 0 | 0 | 0
  DU172.17 at dilution 50, measured at Month 1 | 0 | 0 | 0 | 2 | 0 | 0
  DU172.17 at dilution 80, measured at Month 1 | 0 | 0 | 0 | 0 | 0 | 0
  Du422.1 at dilution 50, measured at Month 1 | 0 | 0 | 0 | 1 | 0 | 0
  Du422.1 at dilution 80, measured at Month 1 | 0 | 0 | 0 | 0 | 0 | 0
  MW965.26 at dilution 50, measured at Month 1 | 0 | 0 | 0 | 1 | 0 | 0
  MW965.26 at dilution 80, measured at Month 1 | 0 | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Magnitude of Serum Neutralizing Antibodies Against Env-pseudotyped Vaccine Strains (Du422.1, Du172.17 and CH505TF) and a Tier 1A Neutralization Phenotype (MW965.26) Assessed 4 Weeks After a Single Vaccination (Part A) or the First Vaccination (Part B)
Description: Neutralizing antibodies against strains of HIV-1 were measured as a function of reductions in Tat-induced luciferase (Luc) reporter gene expression in TZMbl cells. A serum neutralization titer was defined as the serum dilution that reduced relative luminescence units (RLUs) by 50% and 80% (ID50 and ID80) relative to the RLUs in virus control wells (cells + virus only) after subtraction of background RLU (cells only). The assay performed in TZM-bl cells measured neutralization titers against the Env-pseudotyped vaccine strains (Du422.1, Du172.17 and CH505TF) and a virus that exhibits a tier 1A neutralization phenotype (MW965.26).
Time Frame: Measured at Month 1 for both Part A and Part B
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: titer
Groups:
- Part B, Group 5: Vaccine: AdC7-HIVgp140 5 x 10^10 vp at Month 0 and AdC6-HIVgp140 5 x 10^10 vp at Month 3 and CH505TF/GLA-SE 400mg at Month 6
  Control for AdC6-HIVgp140 or AdC7-HIVgp140, Sodium Chloride for Injection, 0.9%. Control for CH505TF gp120/GLA-SE adjuvanted protein: Sodium Chloride for Injection, 0.9%.
Arm/Group | Part A, Group 1: Vaccine | Part A, Group 2: Vaccine | Part A, Group 3: Placebo | Part B, Group 4: Vaccine | Part B, Group 5: Vaccine | Part B, Group 6: Placebo
Number analyzed (Participants) | 4 | 4 | 2 | 10 | 8 | 2
titer
  CH505TF at dilution 50, measured at Month 1 | 5 [5 to 5] | 5 [5 to 7.1] | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5]
  CH505TF at dilution 80, measured at Month 1 | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5]
  DU172.17 at dilution 50, measured at Month 1 | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5]
  DU172.17 at dilution 80, measured at Month 1 | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5]
  Du422.1 at dilution 50, measured at Month 1 | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5]
  Du422.1 at dilution 80, measured at Month 1 | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5]
  MW965.26 at dilution 50, measured at Month 1 | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5]
  MW965.26 at dilution 80, measured at Month 1 | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5]

15. Secondary Outcome: Part B: Response Rate of HIV-specific Serum IgG Binding Antibodies Assessed 4 Weeks After the Second Vaccination
Description: as for outcome 8
Time Frame: Measured at Month 4 for Part B
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Part B, Group 4: Vaccine | Part B, Group 5: Vaccine | Part B, Group 6: Placebo
Number analyzed (Participants) | 9 | 8 | 2
Participants
  1086C_D7gp120.avi/293F measured at Month 4 | 9 | 7 | 0
  1394C9_G1.D11gp120.avi measured at Month 4 | 4 | 2 | 0
  1428_D11gp120.avi/293F measured at Month 4: number analyzed (Participants) | 9 | 7 | 2
  1428_D11gp120.avi/293F measured at Month 4 | 7 | 4 | 0
  1641A7_D11gp120.avi/293F measured at Month 4 | 8 | 6 | 0
  96ZM651.D11gp120.avi measured at Month 4: number analyzed (Participants) | 9 | 7 | 1
  96ZM651.D11gp120.avi measured at Month 4 | 6 | 3 | 0
  CAP210_D11gp120.avi/293F measured at Month 4: number analyzed (Participants) | 9 | 7 | 2
  CAP210_D11gp120.avi/293F measured at Month 4 | 5 | 3 | 0
  CAP45_D11gp120.avi/293F measured at Month 4 | 6 | 3 | 0
  CH0505_CON D7gp120_avi/293F/Mon measured at Month 4: number analyzed (Participants) | 9 | 7 | 2
  CH0505_CON D7gp120_avi/293F/Mon measured at Month 4 | 5 | 2 | 0
  CH505TF D7gp120d371_avi/293F/Mon measured at Month 4: number analyzed (Participants) | 9 | 7 | 2
  CH505TF D7gp120d371_avi/293F/Mon measured at Month 4 | 6 | 2 | 0
  CH505TFD8N156KN160K_avi/293i Mon measured at Month 4: number analyzed (Participants) | 9 | 7 | 1
  CH505TFD8N156KN160K_avi/293i Mon measured at Month 4 | 6 | 3 | 0
  Ce0042_D11gp120.avi/293F measured at Month 4: number analyzed (Participants) | 9 | 7 | 2
  Ce0042_D11gp120.avi/293F measured at Month 4 | 3 | 2 | 0
  Con 6 gp120/B measured at Month 4 | 8 | 6 | 0
  Con S gp140 CFI measured at Month 4 | 9 | 7 | 0
  Du156_D11gp120.avi/293F measured at Month 4 | 9 | 6 | 0
  TV1c8_D11gp120.avi/293F measured at Month 4 | 9 | 7 | 0
  gp41 measured at Month 4: number analyzed (Participants) | 9 | 6 | 2
  gp41 measured at Month 4 | 8 | 5 | 0
  gp70-001428.2.42 V1V2 measured at Month 4: number analyzed (Participants) | 8 | 7 | 2
  gp70-001428.2.42 V1V2 measured at Month 4 | 0 | 1 | 0
  gp70-1012.11.TC21.3257 V1V2 measured at Month 4: number analyzed (Participants) | 8 | 6 | 2
  gp70-1012.11.TC21.3257 V1V2 measured at Month 4 | 2 | 3 | 0
  gp70-1051.12.C22 V1V2 measured at Month 4: number analyzed (Participants) | 8 | 6 | 2
  gp70-1051.12.C22 V1V2 measured at Month 4 | 1 | 4 | 0
  gp70-1394C9G1 V1V2 measured at Month 4: number analyzed (Participants) | 8 | 7 | 2
  gp70-1394C9G1 V1V2 measured at Month 4 | 0 | 3 | 0
  gp70-7060101641 V1V2 measured at Month 4: number analyzed (Participants) | 8 | 7 | 2
  gp70-7060101641 V1V2 measured at Month 4 | 0 | 1 | 0
  gp70-96ZM651.02 V1v2 measured at Month 4: number analyzed (Participants) | 8 | 7 | 2
  gp70-96ZM651.02 V1v2 measured at Month 4 | 2 | 2 | 0
  gp70-BF1266_431a_V1V2 measured at Month 4: number analyzed (Participants) | 8 | 6 | 2
  gp70-BF1266_431a_V1V2 measured at Month 4 | 0 | 2 | 0
  gp70-CAP210.2.00.E8 V1V2 measured at Month 4: number analyzed (Participants) | 8 | 7 | 2
  gp70-CAP210.2.00.E8 V1V2 measured at Month 4 | 0 | 3 | 0
  gp70-CAP45.2.00.G3 V1V2 measured at Month 4: number analyzed (Participants) | 8 | 7 | 2
  gp70-CAP45.2.00.G3 V1V2 measured at Month 4 | 0 | 1 | 0
  gp70-Ce1086_B2 V1V2 measured at Month 4: number analyzed (Participants) | 8 | 7 | 2
  gp70-Ce1086_B2 V1V2 measured at Month 4 | 0 | 1 | 0
  gp70-Ce1176 V1V2 measured at Month 4: number analyzed (Participants) | 8 | 7 | 2
  gp70-Ce1176 V1V2 measured at Month 4 | 0 | 2 | 0
  gp70-Ce704010042_2ES V1V2 measured at Month 4: number analyzed (Participants) | 8 | 7 | 2
  gp70-Ce704010042_2ES V1V2 measured at Month 4 | 0 | 1 | 0
  gp70-ConC V1V2 measured at Month 4: number analyzed (Participants) | 8 | 7 | 2
  gp70-ConC V1V2 measured at Month 4 | 0 | 1 | 0
  gp70-Du156.12 V1V2 measured at Month 4: number analyzed (Participants) | 8 | 7 | 2
  gp70-Du156.12 V1V2 measured at Month 4 | 0 | 1 | 0
  gp70-TV1.21 V1V2 measured at Month 4: number analyzed (Participants) | 8 | 6 | 2
  gp70-TV1.21 V1V2 measured at Month 4 | 0 | 2 | 0
  gp70_CH505TF_V1V2_N156KN160K_avi/293F measured at Month 4: number analyzed (Participants) | 8 | 6 | 1
  gp70_CH505TF_V1V2_N156KN160K_avi/293F measured at Month 4 | 0 | 1 | 0
  gp70_CH505TF_V1V2_avi/293F measured at Month 4: number analyzed (Participants) | 8 | 6 | 1
  gp70_CH505TF_V1V2_avi/293F measured at Month 4 | 0 | 1 | 0

16. Secondary Outcome: Part B: Magnitude of HIV-specific Serum IgG Binding Antibodies Assessed 4 Weeks After the Second Vaccination
Description: as for outcome 9
Time Frame: Measured at Month 4 for Part B
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: Net MFI
Arm/Group | Part B, Group 4: Vaccine | Part B, Group 5: Vaccine | Part B, Group 6: Placebo
Number analyzed (Participants) | 9 | 8 | 2
Net MFI
  1086C_D7gp120.avi/293F measured at Month 4 | 7160.2 [2493 to 22000] | 5318.9 [1591.6 to 22000] | 15.2 [8.1 to 22.4]
  1394C9_G1.D11gp120.avi measured at Month 4 | 287.2 [189.2 to 1066.5] | 168.6 [99.9 to 2388.9] | 1 [1 to 1]
  1428_D11gp120.avi/293F measured at Month 4: number analyzed (Participants) | 9 | 7 | 2
  1428_D11gp120.avi/293F measured at Month 4 | 1886 [1202.5 to 11290] | 1826.8 [453.2 to 12090] | 2131.1 [1066.1 to 3196.2]
  1641A7_D11gp120.avi/293F measured at Month 4 | 2174.2 [1228 to 13183.5] | 2312.1 [673.7 to 22000] | 104.5 [52.8 to 156.2]
  96ZM651.D11gp120.avi measured at Month 4: number analyzed (Participants) | 9 | 7 | 1
  96ZM651.D11gp120.avi measured at Month 4 | 3297.8 [884.5 to 8019] | 844.8 [657.5 to 12190.2] | 1 [1 to 1]
  CAP210_D11gp120.avi/293F measured at Month 4: number analyzed (Participants) | 9 | 7 | 2
  CAP210_D11gp120.avi/293F measured at Month 4 | 1553 [502.5 to 9846.8] | 437.5 [250.4 to 11716] | 3179.5 [1590.2 to 4768.8]
  CAP45_D11gp120.avi/293F measured at Month 4 | 595.5 [386 to 3380.2] | 653.6 [251.8 to 11100.8] | 388.6 [194.8 to 582.4]
  CH0505_CON D7gp120_avi/293F/Mon measured at Month 4: number analyzed (Participants) | 9 | 7 | 2
  CH0505_CON D7gp120_avi/293F/Mon measured at Month 4 | 1790.2 [359.2 to 3655.2] | 355 [242.1 to 11501.5] | 3982.1 [1991.6 to 5972.7]
  CH505TF D7gp120d371_avi/293F/Mon measured at Month 4: number analyzed (Participants) | 9 | 7 | 2
  CH505TF D7gp120d371_avi/293F/Mon measured at Month 4 | 1589.8 [289.5 to 4195.2] | 340.2 [184.2 to 11551.4] | 3744.6 [1872.8 to 5616.4]
  CH505TFD8N156KN160K_avi/293i Mon measured at Month 4: number analyzed (Participants) | 9 | 7 | 1
  CH505TFD8N156KN160K_avi/293i Mon measured at Month 4 | 1826.2 [356 to 3587.5] | 364 [218 to 10714.8] | 1 [1 to 1]
  Ce0042_D11gp120.avi/293F measured at Month 4: number analyzed (Participants) | 9 | 7 | 2
  Ce0042_D11gp120.avi/293F measured at Month 4 | 561.2 [161 to 1006.5] | 207 [174.8 to 4715.1] | 457 [229 to 685]
  Con 6 gp120/B measured at Month 4 | 889 [491.2 to 4699.8] | 979.9 [94.2 to 6685.2] | 27.5 [14.2 to 40.8]
  Con S gp140 CFI measured at Month 4 | 22000 [19531.5 to 22000] | 22000 [22000 to 22000] | 654.1 [337.1 to 971.2]
  Du156_D11gp120.avi/293F measured at Month 4 | 3444.8 [2452.5 to 21158] | 5790.4 [1533.3 to 20619.8] | 84.4 [42.7 to 126.1]
  TV1c8_D11gp120.avi/293F measured at Month 4 | 5688.5 [3846 to 22000] | 9944.1 [1892.9 to 22000] | 197.8 [99.4 to 296.1]
  gp41 measured at Month 4: number analyzed (Participants) | 9 | 6 | 2
  gp41 measured at Month 4 | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 1532.9 [1025.3 to 2040.4]
  gp70-001428.2.42 V1V2 measured at Month 4: number analyzed (Participants) | 8 | 7 | 2
  gp70-001428.2.42 V1V2 measured at Month 4 | 1 [1 to 20.2] | 83.2 [1 to 2134.5] | 1 [1 to 1]
  gp70-1012.11.TC21.3257 V1V2 measured at Month 4: number analyzed (Participants) | 8 | 6 | 2
  gp70-1012.11.TC21.3257 V1V2 measured at Month 4 | 31.5 [1 to 103.9] | 194.2 [98.3 to 676.2] | 13.8 [7.4 to 20.1]
  gp70-1051.12.C22 V1V2 measured at Month 4: number analyzed (Participants) | 8 | 6 | 2
  gp70-1051.12.C22 V1V2 measured at Month 4 | 1 [1 to 34.2] | 295.5 [52.9 to 679.5] | 1 [1 to 1]
  gp70-1394C9G1 V1V2 measured at Month 4: number analyzed (Participants) | 8 | 7 | 2
  gp70-1394C9G1 V1V2 measured at Month 4 | 7.5 [1 to 79.9] | 188.5 [1 to 4973.2] | 1 [1 to 1]
  gp70-7060101641 V1V2 measured at Month 4: number analyzed (Participants) | 8 | 7 | 2
  gp70-7060101641 V1V2 measured at Month 4 | 1 [1 to 9.5] | 1 [1 to 1485] | 1 [1 to 1]
  gp70-96ZM651.02 V1v2 measured at Month 4: number analyzed (Participants) | 8 | 7 | 2
  gp70-96ZM651.02 V1v2 measured at Month 4 | 447 [83.1 to 1022.8] | 609.8 [270.4 to 3245.8] | 1 [1 to 1]
  gp70-BF1266_431a_V1V2 measured at Month 4: number analyzed (Participants) | 8 | 6 | 2
  gp70-BF1266_431a_V1V2 measured at Month 4 | 1 [1 to 97.2] | 107.8 [18.8 to 3505.3] | 1 [1 to 1]
  gp70-CAP210.2.00.E8 V1V2 measured at Month 4: number analyzed (Participants) | 8 | 7 | 2
  gp70-CAP210.2.00.E8 V1V2 measured at Month 4 | 1 [1 to 1] | 167.8 [39.2 to 1172] | 1 [1 to 1]
  gp70-CAP45.2.00.G3 V1V2 measured at Month 4: number analyzed (Participants) | 8 | 7 | 2
  gp70-CAP45.2.00.G3 V1V2 measured at Month 4 | 1 [1 to 5.9] | 84.5 [1 to 1412.5] | 1 [1 to 1]
  gp70-Ce1086_B2 V1V2 measured at Month 4: number analyzed (Participants) | 8 | 7 | 2
  gp70-Ce1086_B2 V1V2 measured at Month 4 | 157.9 [92 to 246.5] | 219.8 [16.6 to 4753.5] | 1 [1 to 1]
  gp70-Ce1176 V1V2 measured at Month 4: number analyzed (Participants) | 8 | 7 | 2
  gp70-Ce1176 V1V2 measured at Month 4 | 1 [1 to 1] | 114.8 [8.4 to 1575.8] | 1 [1 to 1]
  gp70-Ce704010042_2ES V1V2 measured at Month 4: number analyzed (Participants) | 8 | 7 | 2
  gp70-Ce704010042_2ES V1V2 measured at Month 4 | 1 [1 to 1] | 1 [1 to 358.1] | 1 [1 to 1]
  gp70-ConC V1V2 measured at Month 4: number analyzed (Participants) | 8 | 7 | 2
  gp70-ConC V1V2 measured at Month 4 | 1 [1 to 1] | 3 [1 to 1500] | 1 [1 to 1]
  gp70-Du156.12 V1V2 measured at Month 4: number analyzed (Participants) | 8 | 7 | 2
  gp70-Du156.12 V1V2 measured at Month 4 | 1 [1 to 2.7] | 1 [1 to 12.1] | 1 [1 to 1]
  gp70-TV1.21 V1V2 measured at Month 4: number analyzed (Participants) | 8 | 6 | 2
  gp70-TV1.21 V1V2 measured at Month 4 | 42.1 [1 to 59.5] | 331.6 [1 to 3697.9] | 14.2 [7.6 to 20.9]
  gp70_CH505TF_V1V2_N156KN160K_avi/293F measured at Month 4: number analyzed (Participants) | 8 | 6 | 1
  gp70_CH505TF_V1V2_N156KN160K_avi/293F measured at Month 4 | 1 [1 to 1] | 244 [50.2 to 461.6] | 93.8 [93.8 to 93.8]
  gp70_CH505TF_V1V2_avi/293F measured at Month 4: number analyzed (Participants) | 8 | 6 | 1
  gp70_CH505TF_V1V2_avi/293F measured at Month 4 | 1 [1 to 79.7] | 1463 [342.8 to 1770.2] | 307.8 [307.8 to 307.8]

17. Secondary Outcome: Part B: HIV-specific Serum IgG Binding Antibodies Magnitude Breadth of AUC by Panel and Treatment Arm Assessed 4 Weeks After the Second Vaccination
Description: as for outcome 10
Time Frame: Measured at Month 4 for Part B
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: log10(net MFI)
Arm/Group | Part B, Group 4: Vaccine | Part B, Group 5: Vaccine | Part B, Group 6: Placebo
Number analyzed (Participants) | 9 | 8 | 2
log10(net MFI)
  Clade C gp120 measured at Month 4: number analyzed (Participants) | 9 | 7 | 1
  Clade C gp120 measured at Month 4 | 2.94 [2.51 to 3.84] | 2.64 [2.21 to 3.61] | 2 [2 to 2]
  Clade C gp70 V1V2 measured at Month 4: number analyzed (Participants) | 8 | 6 | 2
  Clade C gp70 V1V2 measured at Month 4 | 2 [2 to 2.04] | 2.05 [2.01 to 2.45] | 2 [2 to 2]

18. Secondary Outcome: Part B: Response Rate of HIV-specific CD4+ and CD8+ T-cell Responses Assessed 4 Weeks After the Second Vaccination
Description: as for outcome 11
Time Frame: Measured at Month 4 for Part B
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Part B, Group 4: Vaccine | Part B, Group 5: Vaccine | Part B, Group 6: Placebo
Number analyzed (Participants) | 9 | 8 | 2
Participants
  Any Env for CD4+ T Cells, measured at Month 4 | 3 | 6 | 0
  Any Env for CD8+ T Cells, measured at Month 4 | 5 | 5 | 0
  ENV-1-PTEG-SEQ for CD4+ T Cells, measured at Month 4: number analyzed (Participants) | 8 | 8 | 2
  ENV-1-PTEG-SEQ for CD4+ T Cells, measured at Month 4 | 3 | 6 | 0
  ENV-1-PTEG-SEQ for CD8+ T Cells, measured at Month 4: number analyzed (Participants) | 8 | 8 | 2
  ENV-1-PTEG-SEQ for CD8+ T Cells, measured at Month 4 | 5 | 5 | 0
  ENV-2-PTEG-SEQ for CD4+ T Cells, measured at Month 4 | 3 | 4 | 0
  ENV-2-PTEG-SEQ for CD8+ T Cells, measured at Month 4 | 4 | 5 | 0

19. Secondary Outcome: Part B: Magnitude of HIV-specific CD4+ and CD8+ T-cell by Cytokine, T-cell Subset, Antigen and Treatment Group Assessed 4 Weeks After the Second Vaccination
Description: as for outcome 12
Time Frame: Measured at Month 4 for Part B
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: Percentage of cells
Arm/Group | Part B, Group 4: Vaccine | Part B, Group 5: Vaccine | Part B, Group 6: Placebo
Number analyzed (Participants) | 9 | 8 | 2
Percentage of cells
  Any Env for CD4+ T Cells, measured at Month 4 | 0.049 [0.038 to 0.156] | 0.09 [0.046 to 0.105] | 0.009 [0.008 to 0.009]
  Any Env for CD8+ T Cells, measured at Month 4 | 0.091 [0.012 to 0.154] | 0.11 [0.046 to 0.319] | 0.011 [0.011 to 0.012]
  ENV-1-PTEG-SEQ for CD4+ T Cells, measured at Month 4: number analyzed (Participants) | 8 | 8 | 2
  ENV-1-PTEG-SEQ for CD4+ T Cells, measured at Month 4 | 0.031 [0.019 to 0.052] | 0.046 [0.032 to 0.05] | 0.004 [0.003 to 0.006]
  ENV-1-PTEG-SEQ for CD8+ T Cells, measured at Month 4: number analyzed (Participants) | 8 | 8 | 2
  ENV-1-PTEG-SEQ for CD8+ T Cells, measured at Month 4 | 0.043 [0.011 to 0.081] | 0.074 [0.033 to 0.135] | 0.005 [0.003 to 0.007]
  ENV-2-PTEG-SEQ for CD4+ T Cells, measured at Month 4 | 0.024 [0.019 to 0.108] | 0.04 [0.018 to 0.055] | 0.005 [0.003 to 0.007]
  ENV-2-PTEG-SEQ for CD8+ T Cells, measured at Month 4 | 0.011 [0.006 to 0.074] | 0.03 [0.015 to 0.111] | 0.006 [0.004 to 0.009]

20. Secondary Outcome: Part B: Response Rate of Serum Neutralizing Antibodies Against Env-pseudotyped Vaccine Strains (Du422.1, Du172.17 and CH505TF) and a Tier 1A Neutralization Phenotype (MW965.26) Assessed 4 Weeks After the Second Vaccination
Description: as for outcome 13
Time Frame: Measured at Month 4 for Part B
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Part B, Group 4: Vaccine | Part B, Group 5: Vaccine | Part B, Group 6: Placebo
Number analyzed (Participants) | 9 | 8 | 2
Participants
  CH505TF at dilution 50, measured at Month 4 | 0 | 0 | 1
  CH505TF at dilution 80, measured at Month 4 | 0 | 0 | 0
  DU172.17 at dilution 50, measured at Month 4 | 0 | 0 | 1
  DU172.17 at dilution 80, measured at Month 4 | 0 | 0 | 0
  Du422.1 at dilution 50, measured at Month 4 | 0 | 0 | 1
  Du422.1 at dilution 80, measured at Month 4 | 0 | 0 | 0
  MW965.26 at dilution 50, measured at Month 4 | 8 | 6 | 0
  MW965.26 at dilution 80, measured at Month 4 | 5 | 5 | 0

21. Secondary Outcome: Part B: Magnitude of Serum Neutralizing Antibodies Against Env-pseudotyped Vaccine Strains (Du422.1, Du172.17 and CH505TF) and a Tier 1A Neutralization Phenotype (MW965.26) Assessed 4 Weeks After the Second Vaccination
Description: Neutralizing antibodies against strains of HIV-1 were measured as a function of reductions in Tat-induced luciferase (Luc) reporter gene expression in TZMbl cells. A serum neutralization titer was defined as the serum dilution that reduced relative luminescence units (RLUs) by 50% and 80% (ID50 and ID80) relative to the RLUs in virus control wells (cells + virus only) after subtraction of background RLU (cells only). The assay performed in TZM-bl cells measured neutralization titers against the Env-pseudotyped vaccine strains (Du422.1, Du172.17 and CH505TF) and a virus that exhibits a tier 1A neutralization phenotype (MW965.26).
  A titer was defined as the serum dilution that reduced relative luminescence units (RLUs) by 50% and 80% relative to the RLUs in virus control wells (cells + virus only) after subtraction of background RLU (cells only).
Time Frame: Measured at Month 4 for Part B
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: titer
Arm/Group | Part B, Group 4: Vaccine | Part B, Group 5: Vaccine | Part B, Group 6: Placebo
Number analyzed (Participants) | 9 | 8 | 2
titer
  CH505TF at dilution 50, measured at Month 4 | 5 [5 to 5] | 5 [5 to 5] | 9.5 [7.2 to 11.7]
  CH505TF at dilution 80, measured at Month 4 | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5]
  DU172.17 at dilution 50, measured at Month 4 | 5 [5 to 5] | 5 [5 to 5] | 7.8 [6.4 to 9.2]
  DU172.17 at dilution 80, measured at Month 4 | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5]
  Du422.1 at dilution 50, measured at Month 4 | 5 [5 to 5] | 5 [5 to 5] | 9.9 [7.5 to 12.4]
  Du422.1 at dilution 80, measured at Month 4 | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5]
  MW965.26 at dilution 50, measured at Month 4 | 79.2 [33.8 to 94] | 71 [12.1 to 109.8] | 5 [5 to 5]
  MW965.26 at dilution 80, measured at Month 4 | 14.6 [5 to 32.9] | 14.7 [5 to 23.5] | 5 [5 to 5]

22. Secondary Outcome: Part B: Response Rate of HIV-specific Serum IgG Binding Antibodies Assessed 2 Weeks After the Third Vaccination
Description: as for outcome 8
Time Frame: Measured at Month 6.5 for Part B
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Part B, Group 4: Vaccine | Part B, Group 5: Vaccine | Part B, Group 6: Placebo
Number analyzed (Participants) | 8 | 7 | 2
Participants
  1086C_D7gp120.avi/293F measured at Month 6.5 | 8 | 7 | 0
  1394C9_G1.D11gp120.avi measured at Month 6.5 | 8 | 7 | 0
  1428_D11gp120.avi/293F measured at Month 6.5: number analyzed (Participants) | 8 | 6 | 2
  1428_D11gp120.avi/293F measured at Month 6.5 | 8 | 6 | 0
  1641A7_D11gp120.avi/293F measured at Month 6.5 | 8 | 7 | 0
  96ZM651.D11gp120.avi measured at Month 6.5: number analyzed (Participants) | 8 | 6 | 1
  96ZM651.D11gp120.avi measured at Month 6.5 | 8 | 6 | 0
  CAP210_D11gp120.avi/293F measured at Month 6.5: number analyzed (Participants) | 8 | 6 | 2
  CAP210_D11gp120.avi/293F measured at Month 6.5 | 8 | 6 | 0
  CAP45_D11gp120.avi/293F measured at Month 6.5 | 8 | 7 | 0
  CH0505_CON D7gp120_avi/293F/Mon measured at Month 6.5: number analyzed (Participants) | 8 | 6 | 2
  CH0505_CON D7gp120_avi/293F/Mon measured at Month 6.5 | 8 | 6 | 0
  CH505TF D7gp120d371_avi/293F/Mon measured at Month 6.5: number analyzed (Participants) | 8 | 6 | 2
  CH505TF D7gp120d371_avi/293F/Mon measured at Month 6.5 | 8 | 6 | 0
  CH505TFD8N156KN160K_avi/293i Mon measured at Month 6.5: number analyzed (Participants) | 8 | 6 | 1
  CH505TFD8N156KN160K_avi/293i Mon measured at Month 6.5 | 8 | 6 | 0
  Ce0042_D11gp120.avi/293F measured at Month 6.5: number analyzed (Participants) | 8 | 6 | 2
  Ce0042_D11gp120.avi/293F measured at Month 6.5 | 8 | 6 | 0
  Con 6 gp120/B measured at Month 6.5 | 8 | 7 | 0
  Con S gp140 CFI measured at Month 6.5 | 8 | 7 | 0
  Du156_D11gp120.avi/293F measured at Month 6.5 | 8 | 7 | 0
  TV1c8_D11gp120.avi/293F measured at Month 6.5 | 8 | 7 | 0
  gp41 measured at Month 6.5: number analyzed (Participants) | 8 | 5 | 2
  gp41 measured at Month 6.5 | 7 | 4 | 0
  gp70-001428.2.42 V1V2 measured at Month 6.5: number analyzed (Participants) | 7 | 6 | 2
  gp70-001428.2.42 V1V2 measured at Month 6.5 | 3 | 3 | 0
  gp70-1012.11.TC21.3257 V1V2 measured at Month 6.5: number analyzed (Participants) | 7 | 5 | 2
  gp70-1012.11.TC21.3257 V1V2 measured at Month 6.5 | 4 | 3 | 0
  gp70-1051.12.C22 V1V2 measured at Month 6.5: number analyzed (Participants) | 7 | 5 | 2
  gp70-1051.12.C22 V1V2 measured at Month 6.5 | 3 | 4 | 0
  gp70-1394C9G1 V1V2 measured at Month 6.5: number analyzed (Participants) | 7 | 6 | 2
  gp70-1394C9G1 V1V2 measured at Month 6.5 | 4 | 4 | 0
  gp70-7060101641 V1V2 measured at Month 6.5: number analyzed (Participants) | 7 | 6 | 2
  gp70-7060101641 V1V2 measured at Month 6.5 | 3 | 2 | 0
  gp70-96ZM651.02 V1v2 measured at Month 6.5: number analyzed (Participants) | 7 | 6 | 2
  gp70-96ZM651.02 V1v2 measured at Month 6.5 | 2 | 2 | 0
  gp70-BF1266_431a_V1V2 measured at Month 6.5: number analyzed (Participants) | 7 | 5 | 2
  gp70-BF1266_431a_V1V2 measured at Month 6.5 | 3 | 3 | 0
  gp70-CAP210.2.00.E8 V1V2 measured at Month 6.5: number analyzed (Participants) | 7 | 6 | 2
  gp70-CAP210.2.00.E8 V1V2 measured at Month 6.5 | 2 | 4 | 0
  gp70-CAP45.2.00.G3 V1V2 measured at Month 6.5: number analyzed (Participants) | 7 | 6 | 2
  gp70-CAP45.2.00.G3 V1V2 measured at Month 6.5 | 3 | 2 | 0
  gp70-Ce1086_B2 V1V2 measured at Month 6.5: number analyzed (Participants) | 7 | 6 | 2
  gp70-Ce1086_B2 V1V2 measured at Month 6.5 | 3 | 3 | 0
  gp70-Ce1176 V1V2 measured at Month 6.5: number analyzed (Participants) | 7 | 6 | 2
  gp70-Ce1176 V1V2 measured at Month 6.5 | 1 | 2 | 0
  gp70-Ce704010042_2ES V1V2 measured at Month 6.5: number analyzed (Participants) | 7 | 6 | 2
  gp70-Ce704010042_2ES V1V2 measured at Month 6.5 | 1 | 1 | 0
  gp70-ConC V1V2 measured at Month 6.5: number analyzed (Participants) | 7 | 6 | 2
  gp70-ConC V1V2 measured at Month 6.5 | 2 | 1 | 0
  gp70-Du156.12 V1V2 measured at Month 6.5: number analyzed (Participants) | 7 | 6 | 2
  gp70-Du156.12 V1V2 measured at Month 6.5 | 0 | 1 | 0
  gp70-TV1.21 V1V2 measured at Month 6.5: number analyzed (Participants) | 7 | 5 | 2
  gp70-TV1.21 V1V2 measured at Month 6.5 | 1 | 2 | 0
  gp70_CH505TF_V1V2_N156KN160K_avi/293F measured at Month 6.5: number analyzed (Participants) | 7 | 5 | 1
  gp70_CH505TF_V1V2_N156KN160K_avi/293F measured at Month 6.5 | 2 | 2 | 0
  gp70_CH505TF_V1V2_avi/293F measured at Month 6.5: number analyzed (Participants) | 7 | 5 | 1
  gp70_CH505TF_V1V2_avi/293F measured at Month 6.5 | 3 | 2 | 0

23. Secondary Outcome: Part B: Magnitude of HIV-specific Serum IgG Binding Antibodies Assessed 2 Weeks After the Third Vaccination
Description: as for outcome 9
Time Frame: Measured at Month 6.5 for Part B
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: Net MFI
Arm/Group | Part B, Group 4: Vaccine | Part B, Group 5: Vaccine | Part B, Group 6: Placebo
Number analyzed (Participants) | 8 | 7 | 2
Net MFI
  1086C_D7gp120.avi/293F measured at Month 6.5 | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 13.5 [7.2 to 19.8]
  1394C9_G1.D11gp120.avi measured at Month 6.5 | 20251.9 [4882.5 to 22000] | 5330.2 [3441.4 to 11133.6] | 6 [3.5 to 8.5]
  1428_D11gp120.avi/293F measured at Month 6.5: number analyzed (Participants) | 8 | 6 | 2
  1428_D11gp120.avi/293F measured at Month 6.5 | 22000 [18414.2 to 22000] | 22000 [12803.9 to 22000] | 1499.4 [750.2 to 2248.6]
  1641A7_D11gp120.avi/293F measured at Month 6.5 | 22000 [18493.9 to 22000] | 22000 [15769.4 to 22000] | 70.5 [35.8 to 105.2]
  96ZM651.D11gp120.avi measured at Month 6.5: number analyzed (Participants) | 8 | 6 | 1
  96ZM651.D11gp120.avi measured at Month 6.5 | 22000 [21971.9 to 22000] | 22000 [22000 to 22000] | 1 [1 to 1]
  CAP210_D11gp120.avi/293F measured at Month 6.5: number analyzed (Participants) | 8 | 6 | 2
  CAP210_D11gp120.avi/293F measured at Month 6.5 | 22000 [19094.1 to 22000] | 22000 [14543.1 to 22000] | 2226.2 [1113.6 to 3338.9]
  CAP45_D11gp120.avi/293F measured at Month 6.5 | 22000 [12319.1 to 22000] | 13516.5 [7494 to 22000] | 234.4 [118.9 to 349.8]
  CH0505_CON D7gp120_avi/293F/Mon measured at Month 6.5: number analyzed (Participants) | 8 | 6 | 2
  CH0505_CON D7gp120_avi/293F/Mon measured at Month 6.5 | 22000 [20718.1 to 22000] | 22000 [16872.2 to 22000] | 2943.4 [1472.2 to 4414.6]
  CH505TF D7gp120d371_avi/293F/Mon measured at Month 6.5: number analyzed (Participants) | 8 | 6 | 2
  CH505TF D7gp120d371_avi/293F/Mon measured at Month 6.5 | 22000 [18795.9 to 22000] | 22000 [12295 to 22000] | 2626.6 [1313.8 to 3939.4]
  CH505TFD8N156KN160K_avi/293i Mon measured at Month 6.5: number analyzed (Participants) | 8 | 6 | 1
  CH505TFD8N156KN160K_avi/293i Mon measured at Month 6.5 | 22000 [21365.8 to 22000] | 22000 [17977.8 to 22000] | 1 [1 to 1]
  Ce0042_D11gp120.avi/293F measured at Month 6.5: number analyzed (Participants) | 8 | 6 | 2
  Ce0042_D11gp120.avi/293F measured at Month 6.5 | 22000 [9925.1 to 22000] | 11018.1 [4555.2 to 13940.2] | 314.5 [157.8 to 471.2]
  Con 6 gp120/B measured at Month 6.5 | 22000 [18092.1 to 22000] | 21599.8 [12923.9 to 22000] | 6.9 [3.9 to 9.8]
  Con S gp140 CFI measured at Month 6.5 | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 417.6 [213.3 to 621.9]
  Du156_D11gp120.avi/293F measured at Month 6.5 | 22000 [20249.4 to 22000] | 22000 [20090.5 to 22000] | 55.6 [28.3 to 82.9]
  TV1c8_D11gp120.avi/293F measured at Month 6.5 | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 113.9 [57.4 to 170.3]
  gp41 measured at Month 6.5: number analyzed (Participants) | 8 | 5 | 2
  gp41 measured at Month 6.5 | 11919.2 [9853.8 to 16697.5] | 22000 [22000 to 22000] | 1415.2 [1396.4 to 1434.1]
  gp70-001428.2.42 V1V2 measured at Month 6.5: number analyzed (Participants) | 7 | 6 | 2
  gp70-001428.2.42 V1V2 measured at Month 6.5 | 81.8 [22.5 to 360.5] | 496 [63 to 4034.8] | 1 [1 to 1]
  gp70-1012.11.TC21.3257 V1V2 measured at Month 6.5: number analyzed (Participants) | 7 | 5 | 2
  gp70-1012.11.TC21.3257 V1V2 measured at Month 6.5 | 344 [13.1 to 1232.2] | 601.8 [290.8 to 1328.8] | 1 [1 to 1]
  gp70-1051.12.C22 V1V2 measured at Month 6.5: number analyzed (Participants) | 7 | 5 | 2
  gp70-1051.12.C22 V1V2 measured at Month 6.5 | 283.2 [1 to 635.9] | 399.8 [180.2 to 3368.8] | 1 [1 to 1]
  gp70-1394C9G1 V1V2 measured at Month 6.5: number analyzed (Participants) | 7 | 6 | 2
  gp70-1394C9G1 V1V2 measured at Month 6.5 | 1375.8 [155.2 to 7640] | 1141.5 [135.1 to 10074.1] | 1 [1 to 1]
  gp70-7060101641 V1V2 measured at Month 6.5: number analyzed (Participants) | 7 | 6 | 2
  gp70-7060101641 V1V2 measured at Month 6.5 | 126.5 [1 to 2443.9] | 196.6 [123.2 to 4280.2] | 1.9 [1.4 to 2.3]
  gp70-96ZM651.02 V1v2 measured at Month 6.5: number analyzed (Participants) | 7 | 6 | 2
  gp70-96ZM651.02 V1v2 measured at Month 6.5 | 614.8 [256.6 to 8476.2] | 1780.1 [143.4 to 3878.1] | 1 [1 to 1]
  gp70-BF1266_431a_V1V2 measured at Month 6.5: number analyzed (Participants) | 7 | 5 | 2
  gp70-BF1266_431a_V1V2 measured at Month 6.5 | 1508.5 [19.1 to 1705.4] | 491.2 [228.2 to 9834.2] | 1 [1 to 1]
  gp70-CAP210.2.00.E8 V1V2 measured at Month 6.5: number analyzed (Participants) | 7 | 6 | 2
  gp70-CAP210.2.00.E8 V1V2 measured at Month 6.5 | 1 [1 to 222.8] | 1032.4 [69.9 to 2225.6] | 1 [1 to 1]
  gp70-CAP45.2.00.G3 V1V2 measured at Month 6.5: number analyzed (Participants) | 7 | 6 | 2
  gp70-CAP45.2.00.G3 V1V2 measured at Month 6.5 | 1 [1 to 556.4] | 89.9 [8.2 to 3034.1] | 1 [1 to 1]
  gp70-Ce1086_B2 V1V2 measured at Month 6.5: number analyzed (Participants) | 7 | 6 | 2
  gp70-Ce1086_B2 V1V2 measured at Month 6.5 | 262.5 [88.2 to 6151.6] | 864.4 [325.9 to 9912.2] | 1 [1 to 1]
  gp70-Ce1176 V1V2 measured at Month 6.5: number analyzed (Participants) | 7 | 6 | 2
  gp70-Ce1176 V1V2 measured at Month 6.5 | 1 [1 to 18] | 572.9 [13.6 to 1937.1] | 1 [1 to 1]
  gp70-Ce704010042_2ES V1V2 measured at Month 6.5: number analyzed (Participants) | 7 | 6 | 2
  gp70-Ce704010042_2ES V1V2 measured at Month 6.5 | 1 [1 to 1] | 1 [1 to 2029.6] | 1 [1 to 1]
  gp70-ConC V1V2 measured at Month 6.5: number analyzed (Participants) | 7 | 6 | 2
  gp70-ConC V1V2 measured at Month 6.5 | 66.8 [1 to 163.5] | 161.8 [42.2 to 2484.6] | 1 [1 to 1]
  gp70-Du156.12 V1V2 measured at Month 6.5: number analyzed (Participants) | 7 | 6 | 2
  gp70-Du156.12 V1V2 measured at Month 6.5 | 1 [1 to 1] | 1 [1 to 88.2] | 7.2 [4.1 to 10.4]
  gp70-TV1.21 V1V2 measured at Month 6.5: number analyzed (Participants) | 7 | 5 | 2
  gp70-TV1.21 V1V2 measured at Month 6.5 | 863 [214.1 to 1447] | 694 [278.2 to 7141.5] | 1 [1 to 1]
  gp70_CH505TF_V1V2_N156KN160K_avi/293F measured at Month 6.5: number analyzed (Participants) | 7 | 5 | 1
  gp70_CH505TF_V1V2_N156KN160K_avi/293F measured at Month 6.5 | 623.8 [1 to 2979.4] | 445.8 [423.8 to 1988.2] | 71 [71 to 71]
  gp70_CH505TF_V1V2_avi/293F measured at Month 6.5: number analyzed (Participants) | 7 | 5 | 1
  gp70_CH505TF_V1V2_avi/293F measured at Month 6.5 | 1721.8 [28.9 to 11673.6] | 2548 [1283 to 6476.8] | 286.5 [286.5 to 286.5]

24. Secondary Outcome: Part B: HIV-specific Serum IgG Binding Antibodies Magnitude Breadth of AUC by Panel and Treatment Arm Assessed 2 Weeks After the Third Vaccination
Description: as for outcome 10
Time Frame: Measured at Month 6.5 for Part B
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: log10(net MFI)
Arm/Group | Part B, Group 4: Vaccine | Part B, Group 5: Vaccine | Part B, Group 6: Placebo
Number analyzed (Participants) | 8 | 7 | 2
log10(net MFI)
  Clade C gp120 measured at Month 6.5: number analyzed (Participants) | 8 | 6 | 1
  Clade C gp120 measured at Month 6.5 | 4.34 [4.16 to 4.34] | 4.22 [4.01 to 4.26] | 2 [2 to 2]
  Clade C gp70 V1V2 measured at Month 6.5: number analyzed (Participants) | 7 | 5 | 2
  Clade C gp70 V1V2 measured at Month 6.5 | 2.33 [2.08 to 2.56] | 2.22 [2.08 to 2.9] | 2 [2 to 2]

25. Secondary Outcome: Part B: Response Rate of HIV-specific CD4+ and CD8+ T-cell Responses Assessed 2 Weeks After the Third Vaccination
Description: as for outcome 11
Time Frame: Measured at Month 6.5 for Part B
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Part B, Group 4: Vaccine | Part B, Group 5: Vaccine | Part B, Group 6: Placebo
Number analyzed (Participants) | 8 | 7 | 2
Participants
  Any Env for CD4+ T Cells, measured at Month 6.5 | 7 | 6 | 0
  Any Env for CD8+ T Cells, measured at Month 6.5 | 6 | 5 | 0
  ENV-1-PTEG-SEQ for CD4+ T Cells, measured at Month 6.5 | 7 | 6 | 0
  ENV-1-PTEG-SEQ for CD8+ T Cells, measured at Month 6.5 | 6 | 5 | 0
  ENV-2-PTEG-SEQ for CD4+ T Cells, measured at Month 6.5 | 5 | 6 | 0
  ENV-2-PTEG-SEQ for CD8+ T Cells, measured at Month 6.5 | 3 | 3 | 0

26. Secondary Outcome: Part B: Magnitude of HIV-specific CD4+ and CD8+ T-cell by Cytokine, T-cell Subset, Antigen and Treatment Group Assessed 2 Weeks After the Third Vaccination
Description: as for outcome 12
Time Frame: Measured at Month 6.5 for Part B
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: Percentage of cells
Arm/Group | Part B, Group 4: Vaccine | Part B, Group 5: Vaccine | Part B, Group 6: Placebo
Number analyzed (Participants) | 8 | 7 | 2
Percentage of cells
  Any Env for CD4+ T Cells, measured at Month 6.5 | 0.172 [0.077 to 0.278] | 0.257 [0.119 to 0.313] | 0.007 [0.004 to 0.011]
  Any Env for CD8+ T Cells, measured at Month 6.5 | 0.067 [0.038 to 0.113] | 0.094 [0.041 to 0.25] | 0.002 [0.001 to 0.002]
  ENV-1-PTEG-SEQ for CD4+ T Cells, measured at Month 6.5 | 0.1 [0.068 to 0.166] | 0.158 [0.081 to 0.195] | 0.007 [0.004 to 0.011]
  ENV-1-PTEG-SEQ for CD8+ T Cells, measured at Month 6.5 | 0.059 [0.027 to 0.078] | 0.065 [0.026 to 0.118] | 0.002 [0.001 to 0.002]
  ENV-2-PTEG-SEQ for CD4+ T Cells, measured at Month 6.5 | 0.072 [0.014 to 0.095] | 0.071 [0.051 to 0.132] | 0.001 [0.001 to 0.001]
  ENV-2-PTEG-SEQ for CD8+ T Cells, measured at Month 6.5 | 0.012 [0.007 to 0.036] | 0.03 [0.015 to 0.085] | 0.001 [0.001 to 0.001]

27. Secondary Outcome: Part B: Response Rate of Serum Neutralizing Antibodies Against Env-pseudotyped Vaccine Strains (Du422.1, Du172.17 and CH505TF) and a Tier 1A Neutralization Phenotype (MW965.26) Assessed 2 Weeks After the Third Vaccination
Description: as for outcome 13
Time Frame: Measured at Month 6.5 for Part B
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Part B, Group 4: Vaccine | Part B, Group 5: Vaccine | Part B, Group 6: Placebo
Number analyzed (Participants) | 8 | 7 | 2
Participants
  CH505TF at dilution 50, measured at Month 6.5 | 1 | 2 | 0
  CH505TF at dilution 80, measured at Month 6.5 | 1 | 0 | 0
  DU172.17 at dilution 50, measured at Month 6.5 | 2 | 0 | 0
  DU172.17 at dilution 80, measured at Month 6.5 | 0 | 0 | 0
  Du422.1 at dilution 50, measured at Month 6.5 | 1 | 1 | 0
  Du422.1 at dilution 80, measured at Month 6.5 | 0 | 0 | 0
  MW965.26 at dilution 50, measured at Month 6.5 | 8 | 7 | 0
  MW965.26 at dilution 80, measured at Month 6.5 | 8 | 7 | 0

28. Secondary Outcome: Part B: Magnitude of Serum Neutralizing Antibodies Against Env-pseudotyped Vaccine Strains (Du422.1, Du172.17 and CH505TF) and a Tier 1A Neutralization Phenotype (MW965.26) Assessed 2 Weeks After the Third Vaccination
Description: as for outcome 21
Time Frame: Measured at Month 6.5 for Part B
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: titer
Arm/Group | Part B, Group 4: Vaccine | Part B, Group 5: Vaccine | Part B, Group 6: Placebo
Number analyzed (Participants) | 8 | 7 | 2
titer
  CH505TF at dilution 50, measured at Month 6.5 | 5 [5 to 5] | 5 [5 to 8.2] | 5 [5 to 5]
  CH505TF at dilution 80, measured at Month 6.5 | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5]
  DU172.17 at dilution 50, measured at Month 6.5 | 5 [5 to 7.9] | 5 [5 to 5] | 5 [5 to 5]
  DU172.17 at dilution 80, measured at Month 6.5 | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5]
  Du422.1 at dilution 50, measured at Month 6.5 | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5]
  Du422.1 at dilution 80, measured at Month 6.5 | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5]
  MW965.26 at dilution 50, measured at Month 6.5 | 2298.1 [898.4 to 3121.5] | 418.7 [102.2 to 1335.6] | 5 [5 to 5]
  MW965.26 at dilution 80, measured at Month 6.5 | 757.6 [149 to 1145.8] | 104.5 [31.1 to 350.7] | 5 [5 to 5]

ADVERSE EVENTS:
Time Frame: All adverse events were collected for 30 after any receipt of study vaccination (up to 7 months). All serious adverse events (SAEs), medically attended adverse events (MAAEs), and adverse events of special interest (AESIs) were collected for twelve months following any receipt of study product (up to 18 months). Study vaccinations were given at study Day 0 (Month 0) for Part A (T1, T2, and C3) and at study Days 0 (Month 0), 84 (Month 3) and 168 (Month 6) for Part B (T4, T5, and C6).
Arm/Group | Part A, Group 1: Vaccine | Part A, Group 2: Vaccine | Part A, Group 3: Placebo | Part B, Group 4: Vaccine | Part B, Group 5: Vaccine | Part B, Group 6: Placebo
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/2 | 0/10 | 1/10 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/2 | 0/10 | 1/10 | 0/2
Other Adverse Events (participants affected / at risk) | 1/5 | 1/5 | 1/2 | 7/10 | 3/10 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A, Group 1: Vaccine (N=5) | Part A, Group 2: Vaccine (N=5) | Part A, Group 3: Placebo (N=2) | Part B, Group 4: Vaccine (N=10) | Part B, Group 5: Vaccine (N=10) | Part B, Group 6: Placebo (N=2)
Any Event in SOC (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stab wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A, Group 1: Vaccine (N=5) | Part A, Group 2: Vaccine (N=5) | Part A, Group 3: Placebo (N=2) | Part B, Group 4: Vaccine (N=10) | Part B, Group 5: Vaccine (N=10) | Part B, Group 6: Placebo (N=2)
Any Event in SOC (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Any Event in SOC (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 5 (6) | 1 (1) | 0 (0)
Body tinea (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urethritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Any Event in SOC (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Any Event in SOC (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Any Event in SOC (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Any Event in SOC (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Balanoposthitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol: Protocol Version 1 (2021-02-23): https://cdn.clinicaltrials.gov/large-docs/25/NCT05182125/Prot_000.pdf
  • Study Protocol: Letter of Amendment (2022-11-16): https://cdn.clinicaltrials.gov/large-docs/25/NCT05182125/Prot_002.pdf
  • Statistical Analysis Plan: SAP for safety (2024-07-25): https://cdn.clinicaltrials.gov/large-docs/25/NCT05182125/SAP_001.pdf
  • Statistical Analysis Plan: SAP for immunogenicity (2024-09-11): https://cdn.clinicaltrials.gov/large-docs/25/NCT05182125/SAP_003.pdf